CLINICAL TRIAL: NCT02544217
Title: A Phase I, Randomized, Double Blind, Placebo-controlled, Dose-escalating Clinical Trial With KH176
Brief Title: A Dose-escalating Clinical Trial With KH176
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khondrion BV (Industry)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KH176-101
Record Dates: First submitted 2015-04-19; First posted 2015-09-09 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2016-02

CONDITIONS: MELAS; LHON; Leigh Syndrome; Mitochondrial Disease; Mitochondrial DNA tRNALeu(UUR) m.3243A<G Mutation
MeSH Terms: conditions — MELAS Syndrome; Leigh Disease; Mitochondrial Diseases | interventions — 6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Escalating (Experimental): 2 alternating groups receiving escalating single doses of active/placebo
  Interventions: Drug: KH176; Drug: placebo
- Multiple Escalating (Experimental): 3 multiple escalating groups, receiving active/placebo
  Interventions: Drug: KH176; Drug: placebo

INTERVENTIONS:
Drug: KH176
Drug: placebo

SUMMARY:
Mitochondrial Diseases are rare progressive, multi-system, often early fatal disorders affecting both children and adults. KH176 is a novel chemical entity currently under development for the treatment of inherited mitochondrial diseases, including MELAS (Mitochondrial Encephalomyopathy, Lactic acidosis, and Stroke-like episodes), Leigh's Disease and Leber's Hereditary Optic Neuropathy (LHON). KH176 is a potent intracellular redox modulating agent targeting the reactive oxygen species which are important in the pathogenesis of disorders of mitochondrial oxidative phosphorylation. After demonstrating a favourable safety profile in the pre-clinical testing, the safety, tolerability and pharmacokinetic and pharmacodynamic characteristics of the compound will now be evaluated in healthy male subjects in this trial

ELIGIBILITY:
Inclusion Criteria:

* Healthy as assessed by medical history, physical examination, Vital Signs, Clinical Laboratory, ECG

Exclusion Criteria:

* Allergies,
* Concomitant medication,
* concomitant disease,
* relevant surgery,
* recent blood donation

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Research Unit Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Koene S, Spaans E, Van Bortel L, Van Lancker G, Delafontaine B, Badilini F, Beyrath J, Smeitink J. KH176 under development for rare mitochondrial disease: a first in man randomized controlled clinical trial in healthy male volunteers. Orphanet J Rare Dis. 2017 Oct 16;12(1):163. doi: 10.1186/s13023-017-0715-0. PMID 29037240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All studies were conducted at the Drug Research Unit Ghent. Participants agreed to stay in the Drug Research Unit during the first 24 h after dosing (SAD) and during Day 8 (MAD).
Groups:
- Single Ascending Group I; Single Ascending Group II: 2 alternating groups receiving escalating single doses of active/placebo
  KH176
  placebo
- Multiple Ascending Group III; Multiple Ascending Group IV; Multiple Ascending Group V: 3 multiple escalating groups, receiving active/placebo
  KH176
  placebo
- Placebo: Group receiving placebo
Period: Overall Study
Arm/Group | Single Ascending Group I | Single Ascending Group II | Multiple Ascending Group III | Multiple Ascending Group IV | Multiple Ascending Group V | Placebo
Started | 7 | 7 | 4 | 4 | 4 | 6
Completed | 6 | 6 (Two subjects prematurely withdrew from the study for non-medical reasons and were replaced.) | 4 | 4 | 4 | 6
Not Completed | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: SAD:14 subjects divided in two groups of 7 subjects were included. Two subjects prematurely withdrew from the study after dosing period 2 for non-medical reasons. MAD part:18 subjects divided in 3 groups of 6 subjects were included. Two subjects prematurely withdrew from the study for non-medical reasons and were replaced.
Groups:
- SAD Group I: SAD group I: 10mg, 100mg, 800mg
- SAD Group II: SAD group II: 30mg, 300mg, 2000mg
- MAD Group III: MAD group III:100mg bis in die (BID)
- MAD Group IV: MAD group IV: 200mg BID
- MAD Group V: MAD group V: 400mg BID
- Placebo: Placebo group
- Total: Total of all reporting groups
Arm/Group | SAD Group I | SAD Group II | MAD Group III | MAD Group IV | MAD Group V | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 4 | 4 | 4 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (10.5) | 32.0 (11.3) | 40.8 (13.0) | 34.5 (11.6) | 44.0 (8.2) | 44.7 (9.8) | 40.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 4 | 4 | 4 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 6 | 7 | 4 | 3 | 4 | 5 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 7 | 4 | 4 | 4 | 6 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 7 | 7 | 4 | 4 | 4 | 6 | 32
Height [Mean (Standard Deviation); unit: cm] | 178.07 (6.56) | 176.01 (8.11) | 184.63 (2.81) | 181.75 (5.25) | 175.70 (3.18) | 175.55 (8.25) | 184.0 (4.0)
Weight [Mean (Standard Deviation); unit: kg] | 82.86 (10.56) | 74.29 (12.61) | 89.05 (11.84) | 77.85 (11.96) | 81.10 (4.82) | 72.03 (6.06) | 80.0 (8.0)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.09 (2.51) | 24.01 (4.01) | 26.10 (2.74) | 23.60 (3.82) | 26.28 (1.67) | 23.43 (1.98) | 24.0 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: SAD: Change From Baseline in ECG Results by Timepoint: Corrected QT Interval According to Fridericia's Formula (QTcF)
Description: The baseline ECG recording consists of a triplicate recording (3 recordings of a least 3 complexes within a 5 minute window) prior to dosing on Day 1. For the evaluation of the corrected QT intervals the average of the 3 recordings will be taken as baseline. Other ECG recordings will be singlet (one recording of at least 3 complexes) prior to dosing. QTcF is calculated as the quotient between the QT interval in milliseconds and the cube root of the RR interval in seconds, according to Fridericia's formula.
Time Frame: Baseline, 1, 2, 4, 6, 8, 12, 24 hours, 7 day follow up
Population: The safety analysis set included all subjects who have been assigned treatment and have been administered at least once with placebo or KH176.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Group I Placebo; Group II Placebo: Placebo - single dose
- SAD Group I 10mg: 10mg KH176 - single dose
- SAD Group II 30mg: 30mg KH176 - single dose
- SAD Group I 100mg: 100mg KH176 - single dose
- SAD Group II 300mg: 300mg KH176 - single dose
- SAD Group I 800mg: 800mg KH176 - single dose
- SAD Group II 2000mg: 2000mg KH176 - single dose
- Group I Placebo + Food: Placebo + high calorie/high fat breakfast
- Group I 100mg + Food: 100mg KH176 + high calorie/high fat breakfast
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
msec
  Baseline (Pre-dose Day 1) | 386.2 (17.2) | 395.0 (9.8) | 385.8 (14.8) | 399.3 (8.3) | 390.3 (14.6) | 393.5 (14.2) | 386.5 (10.9) | 385.3 (16.8) | 369.0 (14.1) | 386.5 (13.2)
  Change from baseline (BL)at 1h | 4.0 (2.8) | -2.0 (8.7) | -0.3 (3.8) | -3.5 (6.0) | 0.8 (4.0) | 0.8 (5.7) | 0.3 (7.6) | 28.8 (19.0) | 4.5 (19.1) | 5.8 (2.6)
  Change from BL at 2h | 0.5 (7.9) | -4.0 (6.6) | -1.8 (7.9) | -4.8 (6.1) | -4.8 (3.0) | 1.5 (6.0) | 7.8 (10.0) | 28.5 (14.1) | 2.5 (13.4) | 1.8 (5.3)
  Change from BL at 4h | 6.5 (9.4) | -2.2 (11.4) | -3.8 (3.3) | -4.3 (6.2) | 1.0 (5.7) | 3.8 (12.3) | 3.3 (7.2) | 26.0 (8.7) | 8.5 (17.7) | 0.3 (3.9)
  Change from BL at 6h | 6.2 (3.6) | -2.7 (6.0) | 4.3 (6.3) | -4.0 (7.3) | -1.0 (8.3) | 5.8 (8.1) | 5.5 (2.5) | 26.0 (7.9) | 8.5 (12.0) | 6.0 (5.0)
  Change from BL at 8h | -0.8 (7.3) | -7.2 (4.0) | -5.5 (7.4) | -1.8 (9.2) | 4.3 (10.3) | -1.8 (9.0) | 0.8 (7.5) | 23.3 (12.3) | -2.5 (13.4) | 0.5 (5.4)
  Change from BL at 12h | 1.8 (6.7) | -5.2 (4.8) | -1.8 (2.6) | -7.3 (6.8) | 0.0 (4.7) | 0.0 (8.0) | 8.0 (0.8) | 19.3 (11.1) | 5.5 (7.8) | 3.3 (6.2)
  Change from BL at 24h | 5.3 (12.4) | -7.5 (9.3) | -4.0 (7.3) | -4.8 (5.6) | 0.3 (6.2) | -4.3 (6.5) | 0.3 (9.7) | 11.3 (4.7) | -1.0 (8.5) | -3.8 (4.0)
  Change from BL at FU | -0.3 (12.4) | 2.8 (7.9) | -1.3 (10.8) | 2.8 (8.0) | 2.8 (13.1) | 5.0 (6.1) | -5.0 (3.2) | 3.3 (7.6) | 5.5 (10.6) | 6.5 (13.0)

2. Primary Outcome: Pharmacodynamics of KH176
Description: Change from baseline in biochemistry related to Oxidative Phosphorylation (OXPHOS) (glutathione, lactate); MAD group
Time Frame: Day 1, day 7
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: ratio GSH/GSSG
Groups:
- MAD Group III: MAD group III:100mg BID
- Placebo: Mad group: Placebo
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
ratio GSH/GSSG
  Ox glutathione (GSH)/Red Glutathati(GSSG) Day 1-0h | 872 (532) | 2083 (674) | 2275 (792) | 1584 (491)
  GSH/GSSG Day 7-0h | 919 (196) | 1923 (433) | 1918 (1007) | 1694 (572)
  GSH/GSSG Day 7-3h | 779 (87) | 2045 (338) | 1935 (699) | 1712 (465)
  GSH/GSSG Day 7-6h | 1040 (335) | 2113 (687) | 1993 (863) | 1718 (542)
  GSH/GSSG Day 7-12h | 1361 (606) | 1893 (279) | 1875 (697) | 1680 (657)

3. Primary Outcome: Relationship to Study Drug and Severity of Treatment-emergent Adverse Events
Time Frame: 4 months
Population: as for outcome 1
Measure: Number; unit: TEAE
Groups:
- MAD Group III 200mg: 100mg BID/Day (over 7 days)
- MAD Group IV 400mg: 200mg BID/Day (over 7 days)
- MAD Group V 800mg: 400mg BID/Day (over 7 days)
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food | MAD Group III 200mg | MAD Group IV 400mg | MAD Group V 800mg | Placebo
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4 | 4 | 4 | 4 | 6
TEAE
  TEAE | 5 | 2 | 2 | 5 | 7 | 1 | 0 | 28 | 1 | 1 | 9 | 6 | 14 | 17
  Serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not related TEAE | 4 | 0 | 0 | 2 | 6 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 3
  Unlikely related | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
  Possibly related | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 7 | 4 | 9 | 13
  Related | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 25 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Red Blood Cell Count. SAD Group
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells 10^6/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells 10^6/µL
  Baseline (pre-dose Day 1) | 4.947 (0.488) | 4.933 (0.307) | 4.793 (0.455) | 5.030 (0.458) | 4.953 (0.247) | 5.137 (0.393) | 4.973 (0.141) | 4.623 (0.395) | 5.095 (0.120) | 4.985 (0.343)
  Change from BL at 24h | 0.200 (0.495) | 0.095 (0.260) | 0.063 (0.085) | 0.188 (0.153) | 0.170 (0.250) | 0.065 (0.197) | 0.173 (0.200) | 0.325 (0.185) | 0.185 (0.064) | 0.115 (0.208)
  Change from BL at FU | 0.003 (0.215) | -0.013 (0.149) | 0.185 (0.104) | -0.052 (0.183) | 0.083 (0.127) | -0.147 (0.041) | -0.053 (0.209) | 0.125 (0.182) | -0.150 (0.339) | 0.050 (0.211)

5. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Erythrocyte Sedimentation Rate (SAD Group)
Time Frame: Baseline (pre-dose Day1), 24h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mm/hr
  Baseline | 2.3 (1.4) | 2.8 (2.1) | 1.3 (0.5) | 1.8 (1.0) | 2.0 (1.4) | 3.0 (4.0) | 7.3 (8.5) | 4.0 (3.2) | 5.0 (2.8) | 2.5 (3.0)
  Change from BL at 24h | 0.5 (0.5) | 0.3 (1.0) | 0.0 (0.0) | 1.0 (0.8) | 0.0 (0.8) | 0.3 (1.0) | 0.3 (0.6) | 3.0 (3.6) | -0.5 (0.7) | 1.0 (2.0)
  Change from BL at FU | 0.3 (1.2) | 0.3 (1.5) | 0.8 (1.0) | 0.5 (1.7) | 0.5 (1.7) | 0.0 (0.0) | -2.3 (6.8) | 0.5 (1.0) | 0.0 (0.0) | 0.0 (0.0)

6. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Erythrocyte Sedimentation Rate MAD Group
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mm/hr
  Baseline (pre-dose Day 1) | 4.0 (2.4) | 3.0 (1.8) | 2.0 (1.4) | 2.7 (1.8)
  Change from BL at Day 3 | 2.0 (3.5) | 0.8 (0.5) | 0.5 (0.6) | 0.8 (1.7)
  Change from BL at Day 8 | 4.8 (5.7) | 0.8 (2.2) | 2.5 (1.7) | 0.3 (1.4)
  Change from BL at FU | 5.0 (8.2) | 1.3 (1.3) | 1.0 (0.8) | 2.2 (3.5)

7. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Hematocrit SAD Group
Description: Hematocrit is a measure of the ratio of red blood cells (RBCs) in the blood by volume. Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline (pre-dose Day 1), 24 h postdose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %red cells to the volume of whole blood.
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
%red cells to the volume of whole blood.
  Baseline (pre-dose Day 1) | 43.77 (3.35) | 43.13 (2.79) | 43.10 (3.46) | 44.38 (3.28) | 42.98 (1.41) | 44.35 (2.88) | 44.05 (3.17) | 41.35 (1.68) | 44.35 (2.33) | 42.53 (1.50)
  Change from BL at 24h | 0.53 (1.28) | 0.60 (2.10) | 0.75 (0.91) | 1.95 (1.41) | 1.42 (2.12) | 1.03 (2.11) | 1.33 (1.80) | 2.33 (1.87) | 1.90 (0.28) | 0.68 (1.92)
  Change from BL at FU | -0.43 (1.70) | -0.65 (1.37) | 0.85 (1.45) | -0.93 (1.91) | 0.10 (1.66) | -2.02 (0.54) | -1.15 (2.17) | 0.07 (1.41) | -0.65 (3.04) | 0.55 (2.20)

8. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Mean Corpuscular Haemoglobin. SAD
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24 h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
pg/cell
  Baseline (pre-dose Day 1) | 30.32 (1.83) | 29.70 (0.98) | 30.78 (1.71) | 30.38 (0.49) | 30.00 (1.75) | 29.63 (0.68) | 30.28 (1.26) | 29.80 (1.16) | 30.25 (1.77) | 29.65 (2.13)
  Change from BL at 24h - Day 1 | 0.08 (0.34) | 0.23 (0.59) | 0.17 (0.26) | -0.08 (0.26) | -0.15 (0.13) | -0.60 (0.80) | -0.25 (0.37) | 0.33 (0.41) | 0.25 (0.64) | 0.20 (0.34)
  Change from BL at FU | -0.22 (0.15) | 0.05 (0.46) | -0.28 (0.57) | -0.23 (0.51) | -0.42 (0.37) | -0.28 (0.21) | -0.58 (0.22) | 0.12 (0.39) | -0.15 (0.35) | -0.08 (0.15)

9. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Mean Corpuscular Hemoglobin Concentration - SAD
Description: Erythrocyte mean corpuscular hemoglobin concentration (MCHC) is a measure of the average concentration of hemoglobin per red blood cell. Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline (pre-dose Day 1), 24 h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL RBC
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
g/dL RBC
  Baseline (pre-dose Day 1) | 34.15 (0.34) | 33.98 (1.01) | 34.18 (0.46) | 34.38 (0.84) | 34.53 (0.45) | 34.33 (1.07) | 34.20 (0.65) | 33.25 (0.71) | 34.70 (0.57) | 34.68 (0.99)
  Change from BL at 24h - Day 1 | -0.07 (0.32) | 0.43 (0.42) | 0.00 (0.35) | -0.27 (0.39) | -0.17 (0.15) | -1.05 (0.87) | -0.20 (0.42) | 0.82 (0.29) | 0.10 (0.57) | 0.45 (0.68)
  Change from BL at FU | 0.17 (0.62) | 0.47 (0.42) | 0.27 (0.54) | 0.18 (0.60) | -0.05 (0.64) | 0.30 (0.48) | -0.13 (0.61) | 1.00 (0.12) | -0.60 (0.28) | -0.20 (0.42)

10. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Mean Corpuscular Volume - SAD
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24 h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
fL
  Baseline (pre-dose Day 1) | 88.75 (5.36) | 87.52 (3.71) | 90.15 (5.73) | 88.35 (2.88) | 86.93 (4.75) | 86.42 (2.83) | 88.55 (4.57) | 89.73 (4.24) | 87.10 (6.65) | 85.48 (4.36)
  Change from BL at 24h | 0.45 (0.85) | -0.38 (1.09) | 0.35 (0.37) | 0.48 (0.41) | 0.00 (0.08) | 0.85 (0.73) | -0.27 (0.21) | -1.33 (0.72) | 0.60 (0.28) | -0.55 (0.79)
  Change from BL at FU | -1.10 (1.85) | -1.03 (0.46) | -1.68 (0.90) | -0.92 (1.28) | -1.25 (1.54) | -1.52 (0.69) | -1.45 (1.02) | -2.30 (1.00) | 1.10 (0.28) | 0.20 (0.81)

11. Primary Outcome: MAD: Change From Baseline in ECG Results by Time Point: QTcF
Description: The baseline ECG recording consists of a triplicate recording (3 recordings of a least 3 complexes within a 5 minute window) prior to dosing on Day 1. For the evaluation of the corrected QT intervals the average of the 3 recordings will be taken as baseline. Other ECG recordings will be singlet (one recording of at least 3 complexes) prior to dosing, or around the expected Cmax on Day 1 or 7 for the multiple-dose part.
  QTcF is calculated as the quotient between the QT interval in milliseconds and the cube root of the RR interval in seconds, according to Fridericia's formula.
Time Frame: Baseline, Day1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
msec
  Baseline (Pre-dose Day 1) | 397.3 (18.4) | 384.3 (21.7) | 388.5 (4.7) | 393.0 (18.8)
  Change from BL at 2h - Day 1 | 0.5 (7.5) | 5.5 (8.1) | 7.3 (7.0) | 1.7 (5.3)
  Change from BL at 24h - Day 1 | -4.3 (6.6) | 0.5 (5.7) | 3.3 (13.6) | -4.8 (3.7)
  Change from BL Day 7 at 1h - Day 7 | -1.3 (10.2) | -3.0 (3.3) | -6.5 (8.1) | -2.2 (2.7)
  Change from BL Day 7 at 2h - Day 7 | -3.5 (2.5) | -0.3 (8.2) | -0.8 (3.2) | -0.3 (10.1)
  Change from BL Day 7 at 4h | -7.5 (4.7) | -3.8 (3.5) | -5.8 (7.7) | 3.0 (11.2)
  Change from BL Day 7 BL at 6h - Day 7 | -1.8 (7.3) | 2.0 (4.7) | -7.3 (1.9) | -0.5 (21.0)
  Change from BL Day 7 at 8h - Day 7 | -11.3 (3.2) | -3.8 (6.9) | -11.0 (5.3) | 0.8 (3.9)
  Change from BL Day 7 at 12h - Day 7 | -4.3 (4.6) | -5.0 (3.5) | -10.0 (4.7) | 1.7 (6.0)
  Change from BL at pre-dose Day 2 | -4.3 (6.6) | 0.5 (5.7) | 3.3 (13.6) | -4.8 (3.7)
  Change from BL at pre-dose Day 3 | 0.5 (8.6) | 2.8 (6.4) | 10.5 (17.2) | -7.5 (6.8)
  Change from BL at pre-dose Day 4 | 2.5 (14.6) | 0.5 (13.6) | 7.3 (10.2) | -6.7 (8.4)
  Change from BL at pre-dose Day 5 | 6.0 (13.3) | 2.5 (7.2) | 10.8 (6.7) | -5.3 (7.3)
  Change from BL at pre-dose Day 6 | -1.3 (12.5) | -1.5 (6.2) | 7.8 (8.0) | -8.2 (11.8)
  Change from BL at pre-dose Day 7 | -1.0 (11.9) | 3.0 (9.5) | 13.5 (8.7) | -8.8 (9.2)
  Change from BL at FU | -2.3 (5.0) | 4.0 (6.3) | -0.5 (14.4) | 6.7 (14.1)

12. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: White Blood Cell Count. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells 10^3/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells 10^3/µL
  Baseline (pre-dose Day 1) | 4.435 (0.526) | 4.773 (0.548) | 4.313 (0.418) | 4.863 (0.372) | 4.395 (0.694) | 4.475 (0.733) | 4.853 (0.372) | 5.118 (0.647) | 5.815 (2.072) | 5.535 (1.467)
  Change from BL at 24h | 0.343 (0.525) | -0.057 (0.359) | -0.033 (0.317) | 0.160 (0.329) | 0.257 (0.529) | 0.160 (0.753) | 0.528 (0.324) | 0.655 (0.666) | 0.220 (0.721) | -0.280 (0.555)
  Change from BL at FU | 0.258 (0.309) | -0.203 (0.662) | 0.288 (0.211) | -0.073 (0.367) | 0.395 (0.617) | -0.287 (0.618) | 0.215 (0.266) | -0.320 (0.592) | -0.560 (1.202) | -0.745 (1.535)

13. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Lymphocytes. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells/µL
  Baseline (pre-dose Day 1) | 1570.0 (227.0) | 1748.3 (441.1) | 1655.0 (200.4) | 1862.5 (548.2) | 1485.0 (169.2) | 1570.0 (273.1) | 1550.0 (275.3) | 1497.5 (707.6) | 2260.0 (975.8) | 1640.0 (243.2)
  Change from BL at 24h | -13.3 (223.4) | -16.7 (347.3) | -45.0 (192.8) | -172.5 (227.1) | -27.5 (58.0) | 92.5 (225.6) | 287.5 (353.7) | 37.5 (159.9) | -135.0 (261.6) | -70.0 (177.6)
  Change from BL at FU | 86.7 (265.3) | -45.0 (253.3) | 180.0 (186.5) | -92.5 (315.7) | 127.5 (425.2) | -32.5 (174.6) | 135.0 (294.2) | -7.5 (244.0) | -190.0 (410.1) | -27.5 (125.8)

14. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Neutrophils. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells/µL
  Baseline (pre-dose Day 1) | 2276.7 (551.2) | 2296.7 (658.7) | 2117.5 (369.2) | 2365.0 (820.8) | 2380.0 (679.0) | 2197.5 (835.9) | 2565.0 (462.6) | 2360.0 (438.1) | 2280.0 (169.7) | 3192.5 (1523.9)
  Change from BL at 24h | 356.7 (336.9) | 98.3 (171.2) | 7.5 (196.7) | 410.0 (593.0) | 272.5 (419.1) | 165.0 (335.5) | 285.0 (155.0) | 440.0 (601.5) | 445.0 (459.6) | -122.5 (584.3)
  Change from BL at FU | 205.0 (161.8) | -16.7 (335.4) | 90.0 (183.5) | 107.5 (252.1) | 255.0 (519.0) | -167.5 (480.7) | -12.5 (203.5) | -382.5 (232.9) | -205.0 (445.5) | -557.5 (1326.2)

15. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Hematocrit MAD Group
Description: as for outcome 7
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of red cells to volume of whole blood.
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
% of red cells to volume of whole blood.
  Baseline | 39.93 (1.20) | 43.40 (3.51) | 45.10 (1.33) | 43.30 (1.95)
  Change from BL at Day 3 | 2.67 (1.94) | 1.17 (1.69) | 0.13 (0.45) | 1.70 (1.91)
  Change from BL at Day 8 | 3.30 (1.24) | 1.22 (3.26) | 0.10 (1.22) | 1.93 (2.69)
  Change from BL at FU | 0.92 (1.06) | -0.10 (3.26) | -1.05 (0.64) | -0.75 (2.32)

16. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Eosinophils. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells/µL
  Baseline (pre-dose Day 1) | 115.0 (50.1) | 191.7 (109.4) | 110.0 (49.7) | 137.5 (83.4) | 112.5 (36.9) | 200.0 (78.7) | 245.0 (233.6) | 110.0 (71.6) | 650.0 (792.0) | 152.5 (81.0)
  Change from BL at 24h | -5.0 (16.4) | -50.0 (40.5) | -17.5 (9.6) | -22.5 (42.7) | -15.0 (12.9) | -37.5 (47.9) | -25.0 (33.2) | -25.0 (26.5) | -25.0 (7.1) | -30.0 (47.6)
  Change from BL at FU | -13.3 (16.3) | -58.3 (93.5) | -17.5 (25.0) | -12.5 (43.5) | -2.5 (18.9) | -42.5 (61.3) | 77.5 (201.6) | -20.0 (18.3) | -125.0 (205.1) | -42.5 (42.7)

17. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Thrombocytes. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h, FU (7 days post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells 10^3/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells 10^3/µL
  Baseline (pre-dose Day 1) | 209.5 (45.9) | 204.0 (15.7) | 193.0 (31.9) | 223.0 (21.6) | 215.8 (64.0) | 203.8 (7.0) | 202.3 (54.5) | 160.1 (100.8) | 204.5 (67.2) | 215.8 (55.6)
  Change from BL at 24h | 0.0 (9.7) | 4.8 (6.1) | 8.5 (12.4) | 2.3 (12.8) | 3.8 (20.3) | -14.5 (29.7) | 22.3 (13.5) | 23.0 (22.8) | 4.0 (7.1) | 0.3 (9.0)
  Change from BL at FU | 11.8 (14.0) | 22.5 (15.7) | 23.8 (7.4) | 8.5 (24.3) | 16.3 (14.5) | 7.3 (7.9) | 15.8 (14.3) | 21.5 (22.4) | 1.0 (15.6) | 16.3 (12.5)

18. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Basophils. SAD Group
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value ateach timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells/µL
  Baseline (pre-dose Day 1) | 23.3 (5.2) | 25.0 (10.5) | 15.0 (5.8) | 30.0 (18.3) | 15.0 (10.0) | 32.5 (15.0) | 20.0 (11.5) | 22.5 (5.0) | 65.0 (63.6) | 25.0 (17.3)
  Change from BL at 24h | -5.0 (8.4) | 0.0 (8.9) | 2.5 (5.0) | -7.5 (9.6) | 0.0 (0.0) | -5.0 (10.0) | 2.5 (5.0) | 5.0 (5.8) | -20.0 (14.1) | -2.5 (9.6)
  Change from BL at FU | 0.0 (12.6) | -1.7 (7.5) | 5.0 (5.8) | -5.0 (10.0) | 7.5 (9.6) | -5.0 (12.9) | 20.0 (21.6) | 0.0 (8.2) | -15.0 (21.2) | -2.5 (5.0)

19. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Monocytes. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
cells/µL
  Baseline (pre-dose Day 1) | 445.0 (78.2) | 496.7 (71.7) | 407.5 (79.3) | 455.0 (81.9) | 397.5 (133.0) | 467.5 (98.8) | 462.5 (147.1) | 470.0 (87.6) | 550.0 (70.7) | 512.5 (133.5)
  Change from BL at 24h | 1.7 (46.7) | -81.7 (54.9) | 20.0 (78.3) | -45.0 (19.3) | 20.0 (122.7) | -62.5 (185.5) | -25.0 (112.4) | 2.5 (56.8) | -45.0 (21.2) | -55.0 (70.5)
  Change from BL at FU | -21.7 (91.5) | -78.3 (74.9) | 30.0 (136.4) | -70.0 (94.9) | 5.0 (128.2) | -42.5 (86.6) | 0.0 (94.9) | -47.5 (63.4) | -20.0 (127.3) | -110.0 (128.3)

20. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Mean Corpuscular Volume. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fL
Groups:
- Placebo: MAD Placebo group
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
fL
  Baseline (pre-dose Day 1) | 87.00 (0.62) | 89.32 (2.73) | 86.43 (1.29) | 89.02 (2.93)
  Change from BL at Day 3 | -0.05 (0.40) | 0.52 (1.15) | 0.55 (0.71) | 0.40 (1.08)
  Change from BL at Day 8 | -0.10 (1.30) | -0.43 (0.28) | 0.32 (0.90) | 0.28 (0.95)
  Change from BL at FU | 0.60 (0.74) | -0.55 (0.73) | 1.22 (1.31) | 0.65 (0.77)

21. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Hemoglobin. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
g/dL
  Baseline (pre-dose Day 1) | 13.68 (0.59) | 15.23 (1.38) | 15.68 (0.64) | 14.82 (0.67)
  Change from BL at Day 3 | 1.05 (0.66) | 0.42 (0.74) | 0.17 (0.22) | 0.62 (0.50)
  Change from BL at Day 8 | 1.35 (0.37) | 0.55 (1.22) | 0.27 (0.60) | 0.75 (0.83)
  Change from BL at FU | 0.30 (0.49) | -0.05 (1.11) | -0.38 (0.47) | -0.35 (0.63)

22. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: White Blood Cell Count. MAD
Description: Blood samples were collected from participants at the indicated time points for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each time point are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells 10^3/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells 10^3/µL
  Baseline (pre-dose Day 1) | 5.463 (0.579) | 4.753 (0.410) | 5.378 (1.221) | 4.583 (0.487)
  Change from BL at Day 3 | -0.435 (0.631) | 0.480 (0.787) | 0.895 (0.940) | 0.277 (0.932)
  Change from BL at Day 8 | 0.223 (2.237) | 0.480 (0.252) | 0.795 (0.178) | 0.563 (0.983)
  Change from BL at FU | 0.060 (2.519) | 0.230 (0.870) | 1.340 (0.546) | -0.140 (0.930)

23. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Neutrophils. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells/µL
  Baseline (pre-dose Day 1) | 3077.5 (569.5) | 2602.5 (582.4) | 2935.0 (966.6) | 2483.3 (583.6)
  Change from BL at Day 3 | -567.5 (667.9) | 350.0 (602.4) | 437.5 (505.3) | 81.7 (540.7)
  Change from BL at Day 8 | 105.0 (2079.7) | 312.5 (355.1) | 537.5 (174.6) | 261.0 (634.9)
  Change from BL at FU | 185.0 (2317.4) | 177.5 (827.7) | 1010.0 (622.7) | -75.0 (532.1)

24. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Mean Corpuscular Haemoglobin Concentration. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL RBC
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
g/dL RBC
  Baseline (pre-dose Day 1) | 34.28 (1.08) | 35.05 (0.37) | 34.75 (0.62) | 34.23 (0.37)
  Change from BL at Day 3 | 0.30 (0.22) | 0.05 (0.62) | 0.30 (0.39) | 0.08 (0.48)
  Change from BL at Day 8 | 0.47 (0.43) | 0.25 (0.26) | 0.50 (0.44) | 0.17 (0.38)
  Change from BL at FU | -0.08 (0.33) | 0.00 (0.27) | 0.00 (0.65) | -0.22 (0.44)

25. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Lymphocytes. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells/µL
  Baseline (pre-dose Day 1) | 1627.5 (656.0) | 1498.5 (125.1) | 1750.0 (187.4) | 1508.3 (317.1)
  Change from BL at Day 3 | 87.5 (177.8) | 159.0 (188.6) | 390.0 (297.4) | 215.0 (372.3)
  Change from BL at Day 8 | 12.5 (378.5) | 124.0 (148.8) | 237.5 (208.1) | 283.3 (402.6)
  Change from BL at FU | -55.0 (257.5) | 39.0 (382.3) | 262.5 (220.2) | 5.0 (465.9)

26. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Mean Corpuscular Hemoglobin. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
pg/cell
  Baseline (pre-dose Day 1) | 29.80 (0.91) | 31.33 (1.24) | 30.03 (0.49) | 30.47 (0.97)
  Change from BL at Day 3 | 0.25 (0.13) | 0.23 (0.39) | 0.45 (0.26) | 0.20 (0.25)
  Change from BL at Day 8 | 0.40 (0.40) | 0.12 (0.22) | 0.57 (0.62) | 0.25 (0.33)
  Change from BL at FU | 0.15 (0.47) | -0.20 (0.08) | 0.40 (0.41) | 0.02 (0.25)

27. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Red Blood Cell Count. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells 10^6/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells 10^6/µL
  Baseline (pre-dose Day 1) | 4.588 (0.108) | 4.858 (0.380) | 5.217 (0.138) | 4.873 (0.360)
  Change from BL at Day 3 | 0.313 (0.234) | 0.100 (0.193) | -0.017 (0.060) | 0.167 (0.196)
  Change from BL at Day 8 | 0.385 (0.139) | 0.160 (0.362) | -0.007 (0.144) | 0.198 (0.249)
  Change from BL at FU | 0.075 (0.099) | 0.020 (0.350) | -0.192 (0.145) | -0.120 (0.237)

28. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Eosinophils. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells/µL
  Baseline (pre-dose Day 1) | 212.5 (79.3) | 183.5 (84.6) | 127.5 (45.7) | 141.7 (96.2)
  Change from BL at Day 3 | -40.0 (52.3) | -31.0 (53.2) | 7.5 (20.6) | -28.3 (43.6)
  Change from BL at Day 8 | -47.5 (87.3) | -28.5 (66.0) | -10.0 (27.1) | -22.7 (56.4)
  Change from BL at FU | -27.5 (131.8) | 31.5 (26.5) | -17.5 (27.5) | -45.0 (76.4)

29. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Monocytes. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells/µL
  Baseline (pre-dose Day 1) | 505.0 (44.3) | 424.0 (140.9) | 530.0 (134.9) | 418.3 (61.5)
  Change from BL at Day 3 | 75.0 (151.5) | -11.5 (142.6) | 57.5 (115.0) | 1.7 (64.3)
  Change from BL at Day 8 | 137.5 (374.6) | 76.0 (95.3) | 27.5 (42.7) | 24.3 (53.1)
  Change from BL at FU | -52.5 (176.7) | -21.5 (140.5) | 82.5 (76.8) | -43.3 (85.0)

30. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Thrombocytes. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells 10^3/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells 10^3/µL
  Baseline (pre-dose Day 1) | 207.3 (24.6) | 211.5 (41.2) | 199.8 (25.6) | 206.7 (48.1)
  Change from BL at Day 3 | 15.5 (14.5) | 17.5 (9.5) | 27.5 (8.4) | 17.3 (15.1)
  Change from BL at Day 8 | 44.8 (37.6) | 4.8 (22.3) | 31.3 (13.9) | 29.5 (12.5)
  Change from BL at FU | 63.8 (41.3) | 5.5 (21.9) | 33.8 (20.0) | 21.7 (10.7)

31. Primary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Basophils. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), Day 3, Day 8, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
cells/µL
  Baseline (pre-dose Day 1) | 30.0 (8.2) | 34.0 (10.8) | 20.0 (11.5) | 23.3 (10.3)
  Change from BL at Day 3 | 7.5 (17.1) | 8.5 (17.4) | 2.5 (5.0) | 3.3 (8.2)
  Change from BL at Day 8 | 12.5 (20.6) | -6.5 (17.0) | 5.0 (12.9) | 4.0 (14.7)
  Change from BL at FU | 7.5 (15.0) | 1.0 (6.6) | 2.5 (12.6) | 5.0 (18.7)

32. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Aspartate Aminotransferase. SAD Group
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of clinical chemistry parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
U/L
  Baseline (pre-dose Day 1) | 20.5 (5.9) | 16.8 (2.7) | 19.3 (4.3) | 17.5 (3.8) | 18.3 (9.2) | 20.8 (4.4) | 18.8 (6.1) | 17.0 (2.9) | 19.5 (2.1) | 18.5 (4.8)
  Change from BL at 24h | -2.7 (1.2) | 0.3 (2.1) | -0.5 (1.3) | 1.8 (3.0) | -2.5 (4.7) | -0.3 (1.0) | -1.0 (3.3) | 0.5 (2.5) | -1.0 (2.8) | -1.0 (2.2)
  Change from BL at FU | 0.3 (1.0) | 3.3 (5.8) | 2.8 (6.2) | 4.8 (7.6) | 0.3 (4.9) | 0.5 (7.6) | 1.3 (3.6) | 1.0 (3.7) | 3.5 (6.4) | 0.0 (1.4)

33. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Total Protein. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
g/L
  Baseline (pre-dose Day 1) | 67.5 (4.9) | 65.5 (5.2) | 67.0 (4.1) | 67.3 (2.2) | 65.3 (5.0) | 66.0 (1.8) | 66.3 (3.5) | 66.0 (1.4) | 66.5 (2.1) | 66.3 (5.4)
  Change from BL at 24h | 1.3 (2.7) | 3.7 (3.6) | 1.5 (1.0) | 3.0 (2.4) | 2.8 (4.0) | 6.0 (1.6) | 3.0 (5.0) | 9.3 (4.8) | 2.5 (4.9) | 2.3 (4.6)
  Change from BL at FU | 1.5 (2.9) | 3.3 (3.1) | 4.0 (2.2) | 1.8 (3.9) | 3.3 (1.7) | 0.8 (1.7) | 0.0 (2.2) | 4.8 (3.3) | 1.0 (1.4) | 2.3 (3.2)

34. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Gamma-GT. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
U/L
  Baseline (pre-dose Day 1) | 23.5 (26.7) | 19.0 (14.1) | 24.0 (20.0) | 23.0 (16.2) | 12.0 (6.8) | 17.3 (12.1) | 30.0 (30.8) | 21.3 (17.2) | 29.0 (14.1) | 13.5 (5.1)
  Change from BL at 24h | -0.8 (1.7) | 1.2 (2.1) | 0.0 (0.8) | 0.8 (1.7) | 0.3 (1.3) | 1.3 (0.5) | -0.5 (4.4) | 3.8 (3.1) | 0.0 (2.8) | 0.8 (1.0)
  Change from BL at FU | -4.0 (13.8) | 10.0 (16.1) | -1.3 (4.5) | 13.8 (18.4) | 2.5 (2.4) | 11.3 (20.5) | -7.3 (15.6) | 1.8 (2.5) | 3.5 (3.5) | 1.0 (0.8)

35. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Alkaline Phosphatase. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
U/L
  Baseline (pre-dose Day 1) | 62.0 (18.6) | 64.0 (19.8) | 66.0 (18.5) | 75.0 (32.2) | 66.0 (25.0) | 68.3 (28.0) | 53.3 (10.2) | 49.0 (8.9) | 54.5 (2.1) | 62.3 (21.7)
  Change from BL at 24h | -0.2 (3.0) | 1.7 (3.5) | 1.0 (2.8) | -1.8 (8.1) | 1.0 (4.7) | 3.8 (4.6) | 1.3 (3.6) | 6.8 (3.5) | 2.0 (2.8) | 0.8 (3.6)
  Change from BL at FU | -1.5 (9.0) | 1.7 (6.3) | 1.8 (3.5) | -3.8 (18.2) | 1.5 (3.4) | -1.5 (11.3) | -2.0 (5.4) | 4.3 (1.5) | 2.0 (2.8) | -0.8 (4.9)

36. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Creatinine. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 0.927 (0.058) | 0.768 (0.108) | 0.903 (0.028) | 0.810 (0.091) | 0.838 (0.035) | 0.735 (0.108) | 0.918 (0.043) | 0.838 (0.213) | 0.935 (0.078) | 0.863 (0.024)
  Change from BL at 24h | 0.023 (0.050) | 0.067 (0.033) | 0.080 (0.054) | 0.053 (0.076) | 0.040 (0.041) | 0.115 (0.025) | 0.090 (0.043) | 0.075 (0.112) | 0.015 (0.106) | 0.038 (0.071)
  Change from BL at FU | -0.003 (0.048) | 0.065 (0.048) | 0.012 (0.039) | 0.073 (0.056) | 0.088 (0.068) | 0.063 (0.028) | -0.020 (0.096) | -0.017 (0.085) | -0.080 (0.071) | 0.063 (0.068)

37. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Chloride. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mmol/L
  Baseline (pre-dose Day 1) | 102.7 (2.7) | 104.0 (1.7) | 103.8 (1.7) | 104.0 (0.8) | 102.3 (2.4) | 103.0 (1.4) | 103.3 (1.5) | 103.8 (1.7) | 100.5 (2.1) | 101.5 (2.1)
  Change from BL at 24h | -0.5 (1.4) | -2.5 (1.4) | -1.5 (2.5) | -3.5 (0.6) | 0.0 (1.8) | -2.8 (1.0) | -1.3 (1.0) | -3.5 (1.7) | 2.0 (0.0) | -0.5 (1.3)
  Change from BL at FU | -1.5 (3.5) | -3.2 (2.2) | -2.5 (2.1) | -3.5 (1.3) | -0.8 (2.2) | -2.3 (2.2) | -0.8 (3.5) | -3.0 (0.0) | 3.5 (3.5) | 0.0 (2.7)

38. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Total Bilirubin. SAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 0.82 (0.32) | 0.75 (0.60) | 1.03 (0.83) | 0.68 (0.33) | 1.18 (1.03) | 0.53 (0.13) | 0.63 (0.22) | 0.31 (0.19) | 0.45 (0.21) | 1.10 (1.33)
  Change from BL at 24h | 0.30 (0.26) | 0.12 (0.08) | 0.40 (0.08) | 0.38 (0.13) | -0.00 (0.18) | 0.28 (0.10) | -0.03 (0.15) | 0.31 (0.09) | 0.15 (0.07) | 0.27 (0.17)
  Change from BL at FU | 0.13 (0.42) | -0.02 (0.40) | 0.05 (0.13) | 0.13 (0.13) | -0.18 (0.33) | 0.20 (0.18) | 0.00 (0.29) | 0.21 (0.10) | 0.10 (0.14) | -0.10 (0.56)

39. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Alanine Aminotransferase. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
U/L
  Baseline (pre-dose Day 1) | 20.2 (11.3) | 17.2 (6.9) | 19.3 (3.2) | 20.0 (10.1) | 15.0 (6.9) | 19.3 (6.6) | 22.8 (12.8) | 17.8 (6.8) | 19.0 (1.4) | 15.0 (5.7)
  Change from BL at 24h | -1.2 (2.2) | -0.3 (3.2) | 0.8 (2.9) | -1.3 (3.5) | 1.3 (1.3) | -0.3 (2.8) | -2.0 (3.6) | 0.3 (3.9) | 1.5 (2.1) | 1.5 (1.0)
  Change from BL at FU | -1.0 (4.5) | 5.7 (17.7) | 2.3 (7.8) | 8.3 (18.0) | 1.8 (2.6) | 6.0 (21.5) | -2.3 (5.7) | -1.0 (2.9) | 7.5 (9.2) | 1.8 (2.1)

40. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Creatinine Kinase. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
U/L
  Baseline (pre-dose Day 1) | 118.2 (39.3) | 78.7 (5.9) | 181.8 (59.3) | 78.8 (13.4) | 209.3 (223.6) | 82.3 (28.0) | 68.5 (49.5) | 89.5 (45.4) | 82.5 (89.8) | 81.3 (29.4)
  Change from BL at 24h | -34.3 (23.1) | -14.0 (3.3) | -51.0 (34.6) | -12.8 (1.9) | -97.8 (137.1) | -15.5 (14.1) | -14.0 (23.6) | -14.8 (26.9) | -31.5 (43.1) | -14.8 (8.3)
  Change from BL at FU | 13.0 (43.7) | 16.7 (35.7) | -17.3 (88.6) | 24.5 (39.4) | -110.0 (173.1) | 6.0 (7.5) | 15.8 (16.9) | 7.0 (61.9) | 21.5 (17.7) | 18.0 (31.2)

41. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Urea. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 27.5 (9.3) | 24.7 (4.5) | 30.0 (8.4) | 26.0 (7.3) | 24.0 (2.4) | 25.3 (4.1) | 29.3 (10.6) | 34.8 (7.7) | 38.5 (6.4) | 25.8 (5.7)
  Change from BL at 24h | 0.0 (3.9) | 0.2 (4.4) | -2.5 (5.0) | -0.3 (2.5) | 0.0 (2.8) | -0.5 (5.2) | -1.0 (4.7) | -4.0 (8.6) | -9.0 (1.4) | -0.5 (3.3)
  Change from BL at FU | 1.2 (7.1) | 0.5 (7.7) | -0.8 (3.9) | 2.3 (7.7) | 0.3 (4.5) | -2.3 (7.3) | -0.3 (5.4) | -6.8 (11.8) | -8.0 (4.2) | -1.5 (4.7)

42. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Sodium. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mmol/L
  Baseline (pre-dose Day 1) | 141.8 (1.0) | 142.5 (1.2) | 141.5 (0.6) | 142.8 (1.0) | 141.5 (1.7) | 142.0 (0.8) | 142.3 (1.3) | 143.3 (1.0) | 139.5 (0.7) | 140.5 (1.0)
  Change from BL at 24h | -0.2 (1.6) | -0.7 (0.8) | -0.3 (2.2) | -2.0 (1.4) | -0.8 (2.2) | -1.0 (0.8) | 0.5 (0.6) | -1.3 (1.0) | 2.5 (2.1) | 1.0 (2.6)
  Change from BL at FU | -0.3 (2.4) | -1.8 (2.0) | 0.0 (2.7) | -2.3 (2.2) | 0.8 (1.3) | -2.0 (0.8) | 0.5 (2.4) | -2.8 (1.3) | 4.5 (0.7) | 1.8 (0.5)

43. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Potassium. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mmol/L
  Baseline (pre-dose Day 1) | 4.25 (0.18) | 4.27 (0.18) | 4.25 (0.13) | 4.18 (0.25) | 4.03 (0.19) | 4.33 (0.13) | 4.28 (0.32) | 4.50 (0.18) | 4.00 (0.00) | 4.20 (0.22)
  Change from BL at 24h | 0.17 (0.18) | 0.17 (0.21) | 0.07 (0.31) | 0.23 (0.33) | 0.30 (0.22) | -0.05 (0.26) | 0.12 (0.10) | -0.10 (0.16) | 0.25 (0.07) | 0.15 (0.34)
  Change from BL at FU | 0.25 (0.10) | 0.10 (0.26) | 0.30 (0.22) | 0.20 (0.29) | 0.50 (0.22) | 0.10 (0.27) | 0.08 (0.36) | -0.05 (0.10) | 0.30 (0.14) | 0.33 (0.17)

44. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Phosphate. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mmol/L
  Baseline (pre-dose Day 1) | 1.042 (0.066) | 0.998 (0.122) | 1.120 (0.117) | 1.085 (0.133) | 1.023 (0.081) | 0.983 (0.165) | 1.088 (0.142) | 1.128 (0.193) | 1.410 (0.552) | 1.105 (0.154)
  Change from BL at 24h | 0.033 (0.126) | -0.045 (0.094) | -0.035 (0.169) | -0.133 (0.105) | 0.045 (0.172) | -0.060 (0.111) | 0.032 (0.116) | -0.090 (0.164) | -0.180 (0.999) | -0.015 (0.079)
  Change from BL at FU | -0.020 (0.116) | 0.030 (0.172) | -0.077 (0.126) | -0.018 (0.182) | 0.003 (0.046) | -0.070 (0.153) | -0.090 (0.121) | -0.105 (0.135) | -0.395 (0.205) | -0.080 (0.097)

45. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Calcium (Corrected for Albumin). SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mmol/L
  Baseline (pre-dose Day 1) | 2.380 (0.073) | 2.303 (0.087) | 2.290 (0.114) | 2.288 (0.030) | 2.373 (0.116) | 2.358 (0.069) | 2.353 (0.102) | 2.323 (0.044) | 2.340 (0.000) | 2.360 (0.118)
  Change from BL at 24h | 0.033 (0.045) | 0.095 (0.066) | 0.098 (0.050) | 0.093 (0.028) | 0.058 (0.105) | 0.085 (0.059) | 0.078 (0.075) | 0.148 (0.055) | -0.005 (0.021) | 0.075 (0.088)
  Change from BL at FU | 0.010 (0.041) | 0.062 (0.075) | 0.085 (0.070) | 0.073 (0.098) | 0.042 (0.030) | -0.032 (0.006) | -0.005 (0.033) | 0.090 (0.059) | -0.065 (0.049) | 0.055 (0.039)

46. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Uric Acid. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 5.52 (0.84) | 4.85 (0.84) | 5.75 (0.42) | 4.80 (0.37) | 5.48 (0.82) | 4.75 (0.79) | 5.48 (1.07) | 5.10 (0.96) | 5.45 (0.21) | 5.50 (1.41)
  Change from BL at 24h | -0.25 (0.40) | -0.13 (0.23) | -0.28 (0.25) | -0.20 (0.24) | -0.30 (0.12) | -0.25 (0.24) | -0.20 (0.32) | 0.15 (0.42) | -0.60 (0.28) | -0.28 (0.40)
  Change from BL at FU | 0.28 (0.26) | 0.32 (0.50) | 0.22 (0.79) | 0.40 (0.43) | 0.35 (0.53) | 0.30 (0.08) | 0.18 (0.68) | 0.23 (0.22) | 0.40 (0.28) | 0.33 (0.51)

47. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Triiodothyronine (T3). SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
pg/mL
  Baseline (pre-dose Day 1) | 3.65 (0.35) | 3.23 (0.12) | 3.73 (0.21) | 3.40 (0.22) | 3.48 (0.30) | 3.18 (0.17) | 3.18 (0.17) | 3.33 (0.19) | 3.60 (0.14) | 3.63 (0.41)
  Change from BL at 24h | -0.35 (0.28) | -0.10 (0.24) | -0.22 (0.17) | 0.05 (0.31) | -0.07 (0.10) | -0.23 (0.10) | -0.23 (0.36) | -0.13 (0.15) | -0.40 (0.00) | -0.25 (0.17)
  Change from BL at FU | -0.30 (0.28) | 0.42 (0.23) | -0.23 (0.13) | 0.30 (0.23) | -0.13 (0.17) | 0.50 (0.34) | 0.05 (0.13) | 0.20 (0.08) | -0.30 (0.14) | -0.28 (0.15)

48. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Lipase. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
U/L
  Baseline (pre-dose Day 1) | 31.0 (8.2) | 34.8 (16.2) | 39.0 (9.8) | 29.3 (12.7) | 27.3 (7.5) | 33.0 (9.2) | 30.0 (8.0) | 25.5 (6.2) | 42.0 (14.1) | 31.1 (11.8)
  Change from BL at 24h | -1.5 (3.1) | -7.5 (18.5) | -6.3 (6.8) | -1.8 (2.9) | 1.3 (0.5) | 7.3 (16.5) | -1.3 (3.4) | -4.8 (5.1) | -0.5 (2.1) | -2.5 (5.1)
  Change from BL at FU | -1.0 (2.3) | -1.0 (5.5) | -4.5 (12.4) | 8.0 (27.2) | 1.5 (3.0) | -5.0 (3.7) | -2.0 (6.5) | 9.3 (19.8) | -7.0 (4.2) | -2.5 (3.0)

49. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: (Fasting) Glucose. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 85.0 (7.3) | 86.8 (8.9) | 84.8 (7.4) | 88.5 (12.2) | 77.8 (5.7) | 86.3 (9.4) | 87.0 (4.2) | 95.5 (18.7) | 84.0 (5.7) | 78.8 (3.8)
  Change from BL at 24h | -1.0 (3.2) | 1.2 (5.2) | 2.0 (3.7) | -2.0 (3.2) | 7.0 (4.5) | -1.0 (1.4) | 0.5 (3.1) | -2.3 (1.0) | 4.0 (1.4) | 3.3 (1.9)
  Change from BL at FU | -0.2 (7.0) | 5.5 (6.9) | -0.3 (7.7) | 6.3 (6.7) | 7.3 (6.2) | 0.5 (5.9) | -1.3 (5.4) | -1.5 (1.7) | 2.0 (8.5) | 6.3 (3.8)

50. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Human Serum Albumin. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
g/L
  Baseline (pre-dose Day 1) | 46.2 (3.1) | 45.0 (2.8) | 45.3 (3.9) | 45.0 (1.2) | 45.3 (3.4) | 46.0 (1.4) | 44.0 (1.2) | 44.3 (1.5) | 44.0 (1.4) | 45.8 (3.1)
  Change from BL at 24h | -0.3 (1.2) | 1.7 (1.5) | 0.3 (1.5) | 2.0 (2.6) | 1.5 (3.7) | 3.5 (1.3) | 1.5 (3.1) | 5.3 (2.6) | 0.5 (2.1) | 0.0 (2.7)
  Change from BL at FU | 0.2 (1.8) | 2.0 (1.4) | 2.3 (1.5) | 2.0 (2.8) | 1.0 (1.2) | 0.5 (1.3) | 0.0 (0.8) | 3.5 (2.1) | 0.0 (0.0) | 05 (1.7)

51. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Cholesterol. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 176.0 (47.7) | 151.0 (26.6) | 146.3 (37.5) | 149.0 (38.3) | 146.5 (49.7) | 167.5 (42.3) | 212.8 (48.2) | 174.5 (34.5) | 200.5 (10.6) | 166.5 (28.1)
  Change from BL at 24h | 4.8 (5.5) | 12.5 (10.6) | 5.3 (2.2) | 5.3 (6.4) | 9.5 (14.0) | 19.5 (4.0) | 8.3 (21.0) | 25.0 (12.7) | 12.5 (12.0) | 5.8 (10.7)
  Change from BL at FU | 5.0 (20.4) | 26.3 (27.2) | 25.3 (5.1) | 21.5 (15.5) | 28.3 (17.7) | 24.3 (16.7) | -13.8 (33.7) | 6.8 (5.4) | -2.5 (41.7) | 8.3 (9.3)

52. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: High Density Lipoproteins. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 50.0 (11.1) | 49.8 (8.4) | 45.5 (11.0) | 49.5 (8.9) | 40.0 (4.1) | 54.5 (5.5) | 51.5 (9.6) | 48.0 (13.3) | 47.0 (17.0) | 45.8 (7.3)
  Change from BL at 24h | -2.8 (2.4) | 0.5 (3.1) | 1.0 (1.2) | -2.5 (2.9) | -1.3 (2.1) | 2.8 (2.2) | -3.0 (6.0) | 10.0 (7.3) | 2.5 (7.8) | -0.3 (1.5)
  Change from BL at FU | 1.8 (5.2) | 4.5 (5.0) | 6.3 (4.6) | 3.0 (3.6) | 7.3 (2.6) | 2.8 (5.1) | -3.0 (9.9) | 8.8 (7.4) | -2.0 (7.1) | 1.5 (6.1)

53. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Triglycerides. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 72.8 (19.0) | 88.5 (62.1) | 57.3 (13.0) | 84.5 (46.8) | 72.0 (9.6) | 71.0 (33.6) | 76.3 (15.7) | 117.0 (99.5) | 92.5 (57.3) | 86.3 (20.8)
  Change from BL at 24h | 16.7 (7.2) | 19.0 (17.3) | 10.3 (3.0) | 31.0 (18.1) | 20.3 (16.3) | 22.5 (18.4) | 27.0 (9.5) | -10.3 (46.7) | 1.5 (29.0) | 7.8 (20.2)
  Change from BL at FU | 16.5 (24.5) | 24.5 (58.6) | 30.8 (48.8) | 47.3 (75.3) | 12.5 (19.3) | 37.5 (86.5) | 37.8 (47.1) | -16.5 (48.6) | 43.5 (89.8) | -1.8 (18.6)

54. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Low Density Lipoproteins. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 111.1 (41.9) | 83.5 (24.9) | 88.9 (32.5) | 82.5 (35.3) | 92.3 (46.4) | 98.7 (35.6) | 145.9 (45.7) | 103.1 (40.0) | 134.5 (16.3) | 103.5 (25.7)
  Change from BL at 24h | 4.5 (6.9) | 8.3 (4.6) | 2.9 (3.1) | 1.4 (6.4) | 6.4 (10.3) | 12.8 (2.6) | 5.7 (16.2) | 16.7 (7.8) | 10.0 (9.9) | 4.4 (7.1)
  Change from BL at FU | 0.3 (19.7) | 17.0 (15.6) | 13.3 (10.8) | 9.6 (6.9) | 18.5 (16.4) | 14.2 (6.2) | -17.9 (35.8) | 1.3 (7.7) | -8.5 (30.4) | 7.2 (6.8)

55. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Bicarbonate. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mmol/L
  Baseline (pre-dose Day 1) | 25.68 (1.38) | 25.22 (0.51) | 24.78 (1.09) | 25.85 (0.53) | 24.85 (1.21) | 24.28 (0.33) | 27.05 (0.91) | 26.03 (1.80) | 24.90 (0.71) | 25.93 (0.84)
  Change from BL at 24h | -0.05 (1.15) | 0.28 (1.31) | 1.05 (1.27) | 1.18 (0.90) | 0.40 (0.94) | 2.35 (0.70) | -0.17 (0.94) | 0.05 (1.55) | 1.95 (0.64) | 0.05 (0.39)
  Change from BL at FU | -1.22 (1.38) | 0.97 (1.04) | -0.58 (1.46) | 0.95 (0.88) | -0.15 (0.55) | 1.65 (1.20) | -2.38 (1.64) | -0.20 (1.03) | -0.55 (0.49) | -1.23 (0.30)

56. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Thyroid-stimulating Hormone. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mU/L
  Baseline (pre-dose Day 1) | 1.45 (0.56) | 1.26 (0.64) | 1.14 (0.36) | 1.14 (0.55) | 1.50 (0.97) | 1.55 (0.66) | 1.83 (0.78) | 1.59 (1.03) | 2.57 (2.31) | 1.93 (0.95)
  Change from BL at 24h | -0.20 (0.09) | 0.04 (0.29) | -0.12 (0.22) | -0.03 (0.18) | 0.07 (0.22) | 0.46 (0.52) | 0.05 (0.35) | -0.12 (0.25) | -0.54 (0.65) | -0.42 (0.42)
  Change from BL at FU | 0.08 (0.35) | 0.45 (1.02) | 0.10 (0.22) | 0.77 (0.92) | 0.32 (0.27) | 0.11 (0.58) | 0.17 (0.42) | -0.06 (0.21) | -0.69 (0.73) | -0.10 (0.22)

57. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Thyroxine (T4). SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
ng/dL
  Baseline (pre-dose Day 1) | 1.27 (0.14) | 1.22 (0.16) | 1.30 (0.14) | 1.38 (0.17) | 1.25 (0.10) | 1.08 (0.05) | 1.20 (0.14) | 1.15 (0.06) | 1.35 (0.07) | 1.22 (0.17)
  Change from BL at 24h | -0.05 (0.08) | 0.03 (0.05) | -0.08 (0.10) | -0.08 (0.10) | -0.05 (0.06) | 0.12 (0.05) | 0.05 (0.13) | 0.10 (0.08) | 0.05 (0.07) | 0.03 (0.13)
  Change from BL at FU | 0.03 (0.10) | 0.15 (0.10) | 0.02 (0.22) | 0.05 (0.06) | 0.07 (0.05) | 0.22 (0.05) | 0.05 (0.10) | 0.13 (0.05) | -0.10 (0.14) | 0.10 (0.08)

58. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Timepoint: Lactate. SAD Group
Description: as for outcome 32
Time Frame: Baseline (pre-dose Day 1), 24h post dose, FU (7 days post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
mg/dL
  Baseline (pre-dose Day 1) | 7.98 (2.47) | 7.28 (1.86) | 8.65 (3.20) | 8.23 (2.04) | 8.10 (2.93) | 9.03 (2.08) | 7.53 (0.97) | 8.58 (2.68) | 9.85 (1.34) | 8.33 (1.50)
  Change from BL at 24h | -0.80 (1.83) | 1.40 (2.82) | -2.08 (2.41) | 2.10 (3.81) | -0.50 (1.67) | 0.88 (3.62) | 0.78 (1.75) | 3.25 (1.54) | -1.05 (0.07) | 0.40 (2.22)
  Change from BL at FU | 1.05 (4.59) | 3.80 (3.12) | 2.25 (5.84) | 3.45 (3.45) | 1.93 (6.23) | 0.70 (2.45) | -0.02 (3.40) | 4.33 (3.08) | -0.15 (0.64) | 1.70 (4.59)

59. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Total Protein. MAD Group
Description: as for outcome 4
Time Frame: Baseline (pre-dose Day1), Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
g/L
  Baseline (pre-dose Day 1) | 65.3 (3.8) | 67.3 (4.6) | 63.8 (1.3) | 66.0 (2.1)
  Change from BL at Day 3 | 4.0 (2.4) | 2.3 (1.7) | 2.5 (1.7) | 1.7 (2.3)
  Change from BL at Day 8 | 7.0 (2.9) | 4.3 (4.3) | 6.0 (4.1) | 4.8 (1.7)
  Change from BL at FU | 5.0 (3.4) | 4.8 (4.1) | 4.0 (2.9) | 1.8 (2.0)

60. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Alkaline Phosphatase. MAD Group
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of chemistry parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
U/L
  Baseline (pre-dose Day 1) | 66.0 (16.1) | 67.3 (10.7) | 55.3 (7.3) | 52.3 (9.5)
  Change from BL at Day 3 | 7.3 (6.7) | 2.0 (1.4) | 1.5 (3.9) | 1.8 (1.8)
  Change from BL at Day 8 | 13.0 (9.7) | 5.0 (4.2) | 6.0 (6.4) | 3.3 (1.9)
  Change from BL at FU | 9.0 (13.3) | 10.8 (4.6) | 9.8 (5.2) | 3.3 (4.0)

61. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Aspartate Aminotransferase. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
U/L
  Baseline (pre-dose Day 1) | 20.3 (3.8) | 21.5 (5.7) | 18.5 (0.6) | 23.0 (6.6)
  Change from BL at Day 3 | -2.0 (4.2) | -5.0 (1.4) | -2.5 (1.3) | -1.7 (3.6)
  Change from BL at Day 8 | -1.0 (6.1) | -2.8 (1.9) | -0.3 (2.8) | -1.5 (4.8)
  Change from BL at FU | 1.5 (3.9) | 1.3 (4.6) | 9.8 (16.3) | 2.8 (8.2)

62. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Creatine Kinase. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
U/L
  Baseline (pre-dose Day 1) | 129.5 (62.0) | 192.3 (149.4) | 146.5 (70.8) | 229.8 (156.0)
  Change from BL at Day 3 | -48.5 (40.7) | -68.8 (57.3) | -58.0 (53.3) | -106.5 (115.2)
  Change from BL at Day 8 | -50.8 (49.4) | -83.8 (91.7) | -68.0 (57.7) | -123.5 (144.9)
  Change from BL at FU | 27.0 (23.1) | -7.5 (81.2) | 150.5 (313.3) | 42.2 (153.5)

63. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Gamma GT. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
U/L
  Baseline (pre-dose Day 1) | 15.5 (7.0) | 18.3 (9.2) | 20.5 (14.5) | 21.5 (11.3)
  Change from BL at Day 3 | 0.5 (1.0) | 0.3 (1.3) | 2.0 (2.2) | 0.7 (1.2)
  Change from BL at Day 8 | 0.8 (1.9) | 0.3 (3.0) | 1.8 (2.8) | 0.0 (2.2)
  Change from BL at FU | 1.3 (1.3) | -0.5 (3.1) | 1.8 (2.2) | -0.8 (2.5)

64. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Total Bilirubin. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 0.50 (0.47) | 0.55 (0.13) | 0.63 (0.15) | 0.65 (0.29)
  Change from BL at Day 3 | 0.38 (0.22) | 0.05 (0.13) | 0.20 (0.16) | 0.13 (0.08)
  Change from BL at Day 8 | 0.33 (0.26) | 0.03 (0.21) | 0.18 (0.25) | 0.08 (0.08)
  Change from BL at FU | -0.02 (0.32) | -0.08 (0.21) | 0.08 (0.22) | -0.05 (0.19)

65. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Urea. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 24.8 (3.9) | 28.0 (5.5) | 29.8 (5.1) | 30.2 (3.5)
  Change from BL at Day 3 | 6.0 (2.2) | 2.8 (2.4) | 2.0 (2.6) | 2.5 (3.0)
  Change from BL at Day 8 | 5.8 (6.9) | -0.5 (3.1) | 0.5 (1.3) | -1.0 (4.5)
  Change from BL at FU | 2.3 (8.4) | -0.5 (6.8) | -0.5 (7.1) | -0.3 (6.7)

66. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Creatinine. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 0.910 (0.042) | 0.960 (0.079) | 0.913 (0.067) | 0.897 (0.110)
  Change from BL at Day 3 | 0.095 (0.025) | 0.122 (0.033) | 0.165 (0.031) | 0.057 (0.050)
  Change from BL at Day 8 | 0.005 (0.247) | 0.122 (0.069) | 0.133 (0.082) | 0.053 (0.056)
  Change from BL at FU | 0.008 (0.130) | -0.020 (0.024) | 0.017 (0.043) | 0.007 (0.039)

67. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Sodium. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mmol/L
  Baseline (pre-dose Day 1) | 143.8 (1.0) | 141.3 (0.5) | 141.0 (1.4) | 142.0 (0.9)
  Change from BL at Day 3 | -0.5 (0.6) | -1.5 (0.6) | 0.8 (0.5) | -1.0 (0.6)
  Change from BL at Day 8 | -3.0 (0.8) | 0.8 (0.5) | 1.0 (0.8) | -0.5 (1.4)
  Change from BL at FU | -1.5 (1.0) | -0.3 (2.2) | 2.0 (2.2) | 0.2 (2.1)

68. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Potassium. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mmol/L
  Baseline (pre-dose Day 1) | 4.20 (0.08) | 4.35 (0.19) | 4.40 (0.40) | 4.32 (0.17)
  Change from BL at Day 3 | 0.45 (0.19) | 0.33 (0.37) | 0.10 (0.29) | 0.52 (0.49)
  Change from BL at Day 8 | 0.07 (0.30) | 0.15 (0.39) | 0.25 (0.42) | 0.15 (0.41)
  Change from BL at FU | 0.25 (0.39) | 0.45 (0.31) | 0.25 (0.59) | 0.30 (0.26)

69. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Chloride. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mmol/L
  Baseline (pre-dose Day 1) | 103.8 (2.2) | 101.5 (0.6) | 102.0 (1.8) | 102.2 (1.5)
  Change from BL at Day 3 | -2.5 (0.6) | -2.0 (1.8) | -1.5 (0.6) | -1.5 (0.8)
  Change from BL at Day 8 | -3.5 (1.0) | -2.0 (1.4) | -2.8 (1.0) | -2.2 (2.1)
  Change from BL at FU | -2.0 (0.0) | -2.3 (1.9) | -2.0 (0.8) | -1.3 (1.5)

70. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Calcium (Corrected for Albumin). MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mmol/L
  Baseline (pre-dose Day 1) | 2.278 (0.117) | 2.310 (0.058) | 2.265 (0.024) | 2.323 (0.039)
  Change from BL at Day 3 | 0.105 (0.051) | 0.083 (0.067) | 0.048 (0.068) | 0.068 (0.046)
  Change from BL at Day 8 | 0.127 (0.091) | 0.083 (0.063) | 0.100 (0.095) | 0.088 (0.037)
  Change from BL at FU | 0.087 (0.088) | 0.083 (0.075) | 0.045 (0.082) | 0.055 (0.037)

71. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Uric Acid. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 5.65 (1.67) | 4.93 (0.91) | 5.40 (0.80) | 5.25 (1.14)
  Change from BL at Day 3 | 0.50 (0.56) | 0.58 (0.39) | 0.75 (0.62) | -0.07 (0.31)
  Change from BL at Day 8 | 0.28 (1.14) | -0.02 (0.43) | 0.15 (0.58) | -0.63 (0.52)
  Change from BL at FU | 0.08 (0.92) | 0.55 (0.52) | 0.22 (0.81) | -0.05 (0.42)

72. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Lipase. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
U/L
  Baseline (pre-dose Day 1) | 26.5 (6.1) | 26.5 (3.3) | 32.8 (12.1) | 34.2 (10.3)
  Change from BL at Day 3 | -1.8 (3.1) | 0.0 (1.8) | 26.0 (55.4) | 1.2 (4.4)
  Change from BL at Day 8 | -0.3 (4.1) | 1.3 (7.4) | 50.5 (106.4) | 1.0 (5.1)
  Change from BL at FU | 3.5 (3.3) | 17.3 (24.4) | -2.8 (7.4) | -1.8 (7.6)

73. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Alanine Aminotransferase. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
U/L
  Baseline (pre-dose Day 1) | 25.3 (9.7) | 21.3 (17.4) | 20.5 (6.8) | 22.3 (5.2)
  Change from BL at Day 3 | 0.0 (5.9) | -0.3 (2.2) | -1.3 (0.5) | 2.0 (4.2)
  Change from BL at Day 8 | -1.8 (12.9) | 2.3 (2.6) | 0.3 (5.4) | 2.8 (5.9)
  Change from BL at FU | 1.3 (11.4) | 6.3 (8.3) | 4.8 (7.9) | 2.3 (6.9)

74. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Phosphate. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mmol/L
  Baseline (pre-dose Day 1) | 0.978 (0.094) | 1.033 (0.164) | 0.920 (0.121) | 1.000 (0.162)
  Change from BL at Day 3 | 0.102 (0.033) | 0.003 (0.074) | 0.015 (0.073) | -0.005 (0.111)
  Change from BL at Day 8 | 0.052 (0.116) | 0.000 (0.085) | -0.020 (0.068) | -0.002 (0.113)
  Change from BL at FU | -0.030 (0.131) | -0.010 (0.034) | 0.053 (0.189) | -0.002 (0.190)

75. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Human Serum Albumin. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
g/L
  Baseline (pre-dose Day 1) | 43.3 (2.2) | 45.5 (3.1) | 42.8 (0.5) | 44.7 (1.5)
  Change from BL at Day 3 | 3.3 (2.2) | 3.8 (1.3) | 1.3 (1.0) | 1.5 (2.1)
  Change from BL at Day 8 | 5.3 (2.6) | 3.5 (3.0) | 4.0 (1.8) | 3.8 (1.8)
  Change from BL at FU | 2.8 (2.1) | 3.0 (2.4) | 3.3 (2.1) | 1.7 (1.4)

76. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Fasting Glucose. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 89.0 (5.4) | 85.5 (13.8) | 89.8 (7.5) | 87.2 (10.0)
  Change from BL at Day 3 | -6.8 (4.5) | 2.8 (6.3) | -6.8 (7.9) | 1.5 (2.5)
  Change from BL at Day 8 | -6.5 (7.0) | -9.5 (5.5) | -7.0 (6.1) | -3.5 (7.7)
  Change from BL at FU | -2.2 (1.4) | 2.0 (5.7) | -10.8 (7.8) | 0.0 (7.2)

77. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Cholesterol. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 192.8 (33.5) | 191.0 (11.3) | 203.5 (7.4) | 177.8 (30.7)
  Change from BL at Day 3 | 20.0 (11.5) | 8.8 (9.7) | 13.5 (4.0) | 19.7 (15.3)
  Change from BL at Day 8 | 32.3 (25.3) | 2.5 (20.5) | 13.3 (17.7) | 24.3 (24.4)
  Change from BL at FU | 9.3 (14.2) | 8.0 (22.2) | 9.8 (17.8) | -5.5 (8.6)

78. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Triglycerides. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 140.3 (77.7) | 83.5 (26.3) | 114.0 (74.6) | 90.2 (67.5)
  Change from BL at Day 3 | 14.8 (32.2) | 35.5 (32.7) | 30.5 (30.0) | 14.8 (29.3)
  Change from BL at Day 8 | 17.8 (44.2) | 46.8 (26.9) | 69.0 (42.1) | 28.3 (18.2)
  Change from BL at FU | 16.0 (52.1) | 0.5 (33.5) | 20.3 (56.6) | -8.0 (39.0)

79. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Low Density Lipoproteins. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 114.1 (32.7) | 112.9 (19.0) | 127.0 (18.1) | 93.3 (23.7)
  Change from BL at Day 3 | 17.9 (14.5) | 4.9 (5.2) | 9.0 (7.9) | 18.8 (13.6)
  Change from BL at Day 8 | 33.2 (32.8) | 1.4 (13.8) | 3.5 (20.0) | 25.6 (25.7)
  Change from BL at FU | 8.1 (11.0) | 6.9 (9.6) | -1.5 (20.7) | -1.9 (9.7)

80. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: High Density Lipoproteins. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 51.0 (15.1) | 61.0 (20.1) | 53.5 (20.5) | 66.8 (17.7)
  Change from BL at Day 3 | -1.0 (5.7) | -3.0 (4.8) | -1.5 (5.8) | -2.5 (6.2)
  Change from BL at Day 8 | -5.0 (6.1) | -7.8 (8.6) | -3.5 (11.2) | -7.0 (6.6)
  Change from BL at FU | -2.5 (2.1) | 1.3 (9.9) | 7.5 (12.1) | -2.2 (8.9)

81. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Thyroid-stimulating Hormone. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mU/L
  Baseline (pre-dose Day 1) | 1.41 (0.78) | 1.48 (0.45) | 1.20 (0.36) | 1.58 (0.41)
  Change from BL at Day 3 | 0.11 (0.33) | 0.09 (0.21) | 0.48 (0.54) | 0.25 (0.39)
  Change from BL at Day 8 | 0.28 (0.35) | 0.45 (0.23) | 0.75 (0.52) | 0.85 (0.54)
  Change from BL at FU | 0.16 (0.50) | -0.15 (0.29) | 0.05 (0.48) | 0.05 (0.39)

82. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Trilodothyronine (T3). MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 44 | 4 | 4 | 6
pg/mL
  Baseline (pre-dose Day 1) | 3.35 (0.58) | 3.35 (0.26) | 3.30 (0.14) | 3.08 (0.35)
  Change from BL at Day 3 | -0.05 (0.19) | -0.28 (0.29) | -0.15 (0.19) | -0.15 (0.34)
  Change from BL at Day 8 | -0.32 (0.30) | 0.10 (0.27) | -0.13 (0.22) | -0.05 (0.33)
  Change from BL at FU | 0.30 (0.26) | -0.05 (0.30) | 0.18 (0.29) | 0.18 (0.08)

83. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Thyroxine (T4). MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
ng/dL
  Baseline (pre-dose Day 1) | 1.20 (0.08) | 1.25 (0.06) | 1.20 (0.18) | 1.07 (0.14)
  Change from BL at Day 3 | 0.05 (0.06) | 0.02 (0.05) | 0.05 (0.06) | 0.03 (0.08)
  Change from BL at Day 8 | 0.12 (0.05) | 0.07 (0.10) | 0.23 (0.10) | 0.17 (0.10)
  Change from BL at FU | 0.12 (0.05) | 0.03 (0.10) | 0.12 (0.05) | 0.10 (0.06)

84. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Bicarbonate. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mmol/L
  Baseline (pre-dose Day 1) | 27.53 (0.54) | 25.53 (0.92) | 28.53 (0.59) | 27.23 (0.87)
  Change from BL at Day 3 | -0.38 (0.79) | 2.20 (1.51) | 0.10 (1.55) | 0.03 (1.40)
  Change from BL at Day 8 | -1.10 (1.62) | 1.42 (1.59) | -0.55 (1.72) | 0.47 (1.69)
  Change from BL at FU | -1.18 (0.69) | 1.68 (1.27) | -0.32 (1.78) | -0.27 (1.87)

85. Primary Outcome: Change From Baseline in Chemistry Laboratory Test Results by Time Point: Lactate. MAD Group
Description: as for outcome 60
Time Frame: Baseline, Day 3, Day 8, FU (one week after last dosing)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
mg/dL
  Baseline (pre-dose Day 1) | 8.63 (4.26) | 7.00 (1.82) | 7.23 (1.08) | 9.12 (1.94)
  Change from BL at Day 3 | 0.98 (1.06) | 2.23 (4.01) | 1.18 (1.41) | 5.93 (6.62)
  Change from BL at Day 8 | 3.13 (3.00) | 2.30 (2.08) | 1.83 (1.56) | 1.23 (3.66)
  Change from BL at FU | 2.75 (3.30) | 1.08 (1.49) | 6.63 (4.95) | -0.12 (4.07)

86. Primary Outcome: Phospholipidosis
Description: Change from Day 1 to Day 7 in di-docosahexaenoyl (22:6)-bis(monoacylglycerol) phosphate (di-22:6-BMP) and normalized di-22:6-BMP (urine) - MAD
Time Frame: Day 1, Day 7
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
ng/mL
  di-22:6-BMP: Change from Day 1 to Day 7 | -1.473 (4.520) | -3.465 (4.870) | -2.630 (2.633) | -1.592 (3.283)
  Normalized di-22:6-BMP: Change from Day 1 to Day 7 | 1.298 (0.819) | 0.060 (1.152) | 0.337 (1.120) | 1.780 (1.874)

87. Primary Outcome: MAD: Change From Baseline in ECG Results by Time Point: Corrected QT Interval According to Barret's Formaula (QTcB)
Description: The baseline ECG recording consists of a triplicate recording (3 recordings of a least 3 complexes within a 5 minute window) prior to dosing on Day 1. For the evaluation the average of the 3 recordings will be taken as baseline. Other ECG recordings will be singlet (one recording of at least 3 complexes) prior to dosing, or around the expected Cmax on Day 1 or 7 for the multiple- dose part.
Time Frame: Baseline (pre-dose Day 1), Day1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Follow-up
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
msec
  Baseline (Pre-dose Day 1) | 391.3 (10.8) | 381.0 (28.9) | 384.0 (11.0) | 385.2 (15.4)
  Change from baseline at 2h - Day 1 | 3.8 (10.3) | 12.3 (8.8) | 11.8 (9.7) | 0.7 (6.9)
  Change from BL at 24h - Day 1 | -1.0 (9.8) | 0.3 (6.2) | 11.5 (19.2) | -5.7 (9.7)
  Baseline (pre-dose Day 7) | 398.3 (7.9) | 386.5 (26.1) | 402.0 (6.6) | 378.8 (13.3)
  Change from pre-dose Day 7 at 1h - Day 7 | -3.8 (9.1) | -3.8 (7.9) | -10.3 (11.1) | -3.5 (6.0)
  Change from pre-dose Day 7 at 2h - Day 7 | -5.0 (4.2) | 5.8 (15.2) | 2.5 (8.7) | 1.0 (16.2)
  Change from pre-dose Day 7 at 4h | -7.8 (7.7) | -3.8 (6.2) | -6.5 (13.9) | -0.5 (12.1)
  Change from pre-dose Day 7 BL at 6h - Day 7 | 5.3 (9.8) | 12.5 (7.0) | -1.8 (8.3) | 5.8 (23.5)
  Change from pre-dose Day 7 at 8h - Day 7 | -7.0 (2.8) | -4.5 (9.7) | -11.5 (7.2) | 3.0 (6.9)
  Change from pre-dose Day 7 at 12h - Day 7 | 4.5 (11.4) | 3.0 (5.0) | -9.0 (8.1) | 6.7 (5.7)
  Change from BL at pre-dose Day 2 | -1.0 (9.8) | 0.3 (6.2) | 11.5 (19.2) | -5.7 (9.7)
  Change from BL at pre-dose Day 3 | 6.0 (14.1) | 0.5 (9.7) | 20.5 (22.3) | -8.5 (5.8)
  Change from BL at pre-dose Day 4 | 6.5 (11.5) | 2.0 (14.7) | 7.5 (17.1) | -10.2 (5.0)
  Change from BL at pre-dose Day 5 | 13.8 (14.3) | 10.3 (4.3) | 14.0 (14.2) | -8.5 (5.6)
  Change from BL at pre-dose Day 6 | 5.5 (9.9) | -2.3 (6.7) | 13.5 (13.8) | -10.5 (14.5)
  Change from BL at pre-dose Day 7 | 7.0 (6.5) | 5.5 (9.6) | 18.0 (9.2) | -11.3 (7.7)
  Change from BL at FU | 7.8 (9.7) | 11.0 (3.2) | 10.5 (24.4) | 3.8 (14.3)

88. Primary Outcome: MAD: Change From Baseline in ECG Results by Time Point: P Wave-Q Wave Interval (PQ Interval)
Description: The baseline ECG recording consists of a triplicate recording (3 recordings of a least 3 complexes within a 5 minute window) prior to dosing on Day 1. For the evaluation of the PQ interval the average of the 3 recordings will be taken as baseline.
Time Frame: Baseline (pre-dose Day 1), Day1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Follow-up
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Placebo: MAD group:Placebo
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
msec
  Baseline (Pre-dose Day 1) | 185.8 (33.4) | 160.5 (18.5) | 162.0 (7.0) | 171.8 (20.0)
  Change from baseline at 2h - Day 1 | 2.8 (2.8) | -1.5 (3.0) | 6.0 (5.0) | 6.2 (10.3)
  Change from BL at 24h - Day 1 | -5.8 (6.1) | -0.5 (1.9) | 2.0 (6.6) | -6.5 (14.0)
  Baseline (pre-dose Day 7) | 191.5 (33.4) | 164.0 (22.9) | 167.5 (5.3) | 178.3 (11.8)
  Change from pre-dose Day 7 at 1h - Day 7 | -1.0 (4.8) | 5.5 (30) | 6.5 (2.5) | -1.7 (2.0)
  Change from pre-dose Day 7 at 2h - Day 7 | -3.5 (5.7) | -1.5 (3.4) | 4.0 (4.3) | -14.7 (14.7)
  Change from pre-dose Day 7 at 4h | -9.0 (9.0) | -1.0 (3.8) | 0.0 (1.6) | -14.3 (15.0)
  Change from pre-dose Day 7 BL at 6h - Day 7 | -13.0 (4.8) | -3.5 (8.2) | -4.5 (2.5) | -6.7 (5.2)
  Change from pre-dose Day 7 at 8h - Day 7 | -10.0 (5.9) | 0.0 (7.3) | -5.0 (2.6) | -11.3 (4.1)
  Change from pre-dose Day 7 at 12h - Day 7 | -24.0 (23.6) | -1.5 (5.7) | -4.5 (4.1) | -4.0 (7.6)
  Change from BL at pre-dose Day 2 | -5.8 (6.1) | -0.5 (1.9) | 2.0 (6.6) | -6.5 (14.0)
  Change from BL at pre-dose Day 3 | 6.3 (5.4) | 4.5 (2.5) | 0.0 (6.8) | -6.8 (7.3)
  Change from BL at pre-dose Day 4 | 6.3 (3.3) | 9.5 (1.0) | 7.5 (6.8) | -3.8 (19.7)
  Change from BL at pre-dose Day 5 | -2.3 (7.4) | 4.0 (6.2) | 8.5 (10.1) | -2.2 (16.9)
  Change from BL at pre-dose Day 6 | -0.3 (9.5) | 3.0 (4.3) | 6.0 (3.5) | 5.2 (19.0)
  Change from BL at pre-dose Day 7 | 5.8 (6.8) | 3.5 (5.7) | 5.5 (5.7) | 6.5 (20.9)
  Change from BL at FU | -6.8 (12.0) | -2.5 (3.4) | -3.5 (6.4) | 0.5 (16.2)

89. Primary Outcome: MAD: Change From Baseline in ECG Results by Time Point: the Interval That Denotes Depolarization of the Ventricles, Between the Beginning of the Q Wave and the End of the S Wave (QRS Interval)
Description: as for outcome 87
Time Frame: Baseline (pre-dose Day 1), Day1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Follow-up
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
msec
  Baseline (Pre-dose Day 1) | 99.3 (6.9) | 92.5 (6.1) | 85.5 (8.3) | 98.5 (8.2)
  Change from BL at 2h - Day 1 | 1.3 (1.0) | 2.0 (1.4) | 6.0 (2.9) | -0.2 (1.8)
  Change from BL at 24h - Day 1 | 0.3 (2.1) | 2.5 (2.4) | 3.5 (2.6) | -0.8 (1.3)
  Baseline (pre-dose Day 7) | 99.5 (7.2) | 97.0 (5.3) | 87.5 (7.2) | 98.7 (8.8)
  Change from BL Day 7 at 1h - Day 7 | 0.5 (3.0) | 0.0 (2.8) | 5.0 (2.0) | -0.3 (0.8)
  Change from BL Day 7 at 2h - Day 7 | 0.5 (1.9) | 1.0 (1.2) | 5.5 (1.9) | 0.7 (2.4)
  Change from BL Day 7 at 4h | 0.0 (2.8) | -0.5 (1.0) | 2.5 (2.5) | 0.7 (3.0)
  Change from BL Day 7 BL at 6h - Day 7 | 0.5 (1.9) | -2.5 (2.5) | 3.0 (2.0) | 0.7 (2.4)
  Change from BL Day 7 at 8h - Day 7 | -3.5 (1.9) | -0.5 (1.9) | 2.0 (1.6) | 0.7 (4.8)
  Change from BL Day 7 at 12h - Day 7 | -1.5 (3.0) | -2.0 (1.6) | 2.0 (0.0) | -2.0 (3.6)
  Change from BL at pre-dose Day 2 | 0.3 (2.1) | 2.5 (2.4) | 3.5 (2.6) | -0.8 (1.3)
  Change from BL at pre-dose Day 3 | 0.3 (2.1) | 2.5 (1.3) | 2.0 (3.7) | -0.8 (2.4)
  Change from BL at pre-dose Day 4 | -0.8 (1.5) | 5.0 (3.4) | 3.5 (1.7) | -0.5 (2.7)
  Change from BL at pre-dose Day 5 | -0.8 (1.5) | 2.5 (0.6) | 2.5 (1.7) | -0.5 (2.7)
  Change from BL at pre-dose Day 6 | -0.3 (1.3) | 2.0 (2.4) | 1.0 (2.2) | -1.8 (2.0)
  Change from BL at pre-dose Day 7 | 0.3 (0.5) | 4.5 (1.3) | 2.0 (1.4) | 0.2 (3.1)
  Change from BL at FU | 0.3 (2.6) | 0.5 (1.7) | -2.5 (2.4) | -1.8 (5.2)

90. Primary Outcome: MAD: Change From Baseline in ECG Results by Time Point: QT Interval
Description: as for outcome 87
Time Frame: Baseline (pre-dose Day 1), Day1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Follow-up
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MAD Group III | MAD Group IV | MAD Group V | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 6
msec
  Baseline (Pre-dose Day 1) | 410.5 (41.8) | 391.5 (8.5) | 399.0 (11.2) | 410.2 (33.0)
  Change from BL at 2h - Day 1 | -5.5 (10.5) | -7.5 (16.0) | -4.0 (3.7) | 4.2 (10.1)
  Change from BL at 24h - Day 1 | -10.0 (11.9) | 1.0 (8.8) | -14.5 (4.8) | -4.2 (14.6)
  Baseline (pre-dose Day 7) | 393.0 (42.6) | 388.5 (20.6) | 402.0 (18.8) | 406.0 (22.9)
  Change from pre-dose Day 7 at 1h - Day 7 | 5.0 (12.4) | -1.0 (7.4) | 0.0 (9.1) | 1.0 (8.1)
  Change from pre-dose Day 7 at 2h - Day 7 | 0.0 (6.5) | -10.5 (15.4) | -7.5 (10.0) | -2.3 (14.2)
  Change from pre-dose Day 7 at 4h | -7.0 (1.2) | -2.0 (7.1) | -4.0 (11.9) | 10.7 (15.9)
  Change from pre-dose Day 7 BL at 6h - Day 7 | -15.5 (14.2) | -17.0 (15.2) | -16.5 (10.6) | -14.3 (26.8)
  Change from pre-dose Day 7 at 8h - Day 7 | -18.5 (13.7) | -1.0 (12.7) | -11.0 (11.9) | -3.0 (17.9)
  Change from pre-dose Day 7 at 12h - Day 7 | -20.0 (14.1) | -20.0 (6.3) | -11.5 (9.6) | -8.7 (19.9)
  Change from BL at pre-dose Day 2 | -10.0 (11.9) | 1.0 (8.8) | -14.5 (4.8) | -4.2 (14.6)
  Change from BL at pre-dose Day 3 | -10.5 (20.0) | 7.5 (6.6) | -10.0 (9.6) | -6.2 (12.6)
  Change from BL at pre-dose Day 4 | -6.0 (26.1) | -3.5 (13.4) | 6.0 (4.5) | -0.2 (20.7)
  Change from BL at pre-dose Day 5 | -9.0 (24.9) | -13.0 (11.9) | 3.0 (9.4) | 1.2 (16.1)
  Change from BL at pre-dose Day 6 | -16.0 (23.5) | -0.5 (12.2) | -4.5 (10.1) | -3.8 (11.9)
  Change from BL at pre-dose Day 7 | -17.5 (32.3) | -3.0 (14.8) | 3.0 (9.4) | -4.2 (16.1)
  Change from BL at FU | -22.0 (13.2) | -10.5 (14.6) | -23.0 (14.3) | 13.2 (23.9)

91. Primary Outcome: SAD: Change From Baseline in ECG Results by Time Point: PQ Interval
Description: The baseline ECG recording consists of a triplicate recording (3 recordings of a least 3 complexes within a 5 minute window) prior to dosing on Day 1. For the evaluation the average of the 3 recordings will be taken as baseline.
Time Frame: Pre-dose, Day 1, Day 7
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: msec
Groups:
- SAD Group I Placebo: SAD group I - Placebo
- SAD Group II Placebo: SAD group II - Placebo
- Group I Placebo + Food: Placebo - single dose + Food
- Group II 100mg + Food: 100mg KH176 - single dose + Food
Arm/Group | SAD Group I Placebo | SAD Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group II 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
msec
  Baseline (Pre-dose Day 1) | 195.5 (28.9) | 165.0 (21.6) | 154.5 (39.2) | 159.8 (23.0) | 155.0 (24.4) | 176.5 (21.4) | 171.8 (15.9) | 176.0 (17.7) | 177.0 (26.9) | 147.5 (25.2)
  Change from baseline at 1h | -1.2 (4.0) | 3.3 (7.4) | -0.5 (1.9) | -1.3 (5.7) | -4.0 (3.7) | 4.0 (2.8) | 8.8 (3.0) | 20.5 (7.5) | -9.0 (9.9) | -3.5 (4.4)
  Change from BL at 2h post dose | 1.2 (3.9) | -0.7 (3.7) | -3.0 (3.7) | 1.3 (3.8) | -3.0 (3.8) | 4.5 (5.7) | 8.3 (11.8) | 16.0 (5.9) | -11.0 (9.9) | -1.0 (2.6)
  Change from BL at 4h post dose | -1.5 (8.8) | -2.3 (0.8) | -2.0 (2.6) | 4.8 (4.4) | -3.5 (5.3) | 0.0 (4.0) | 3.3 (5.7) | 10.0 (6.3) | -5.0 (7.1) | -1.5 (3.0)
  Change from BL at 6h post dose | -1.2 (3.6) | -2.7 (3.3) | -2.0 (2.6) | 0.8 (7.2) | -7.5 (5.3) | -5.5 (8.5) | -3.3 (8.8) | 9.0 (6.0) | -11.0 (12.7) | -1.5 (1.9)
  Change from BL at 8h post dose | -3.2 (3.6) | 1.0 (6.2) | -6.5 (5.5) | -1.3 (7.4) | -8.0 (4.3) | -8.0 (8.6) | -5.3 (7.8) | 1.0 (10.4) | -6.0 (2.8) | -4.0 (3.7)
  Change from BLat 12h post dose | -1.8 (4.7) | -3.7 (8.3) | -4.0 (4.8) | -1.8 (4.9) | -6.5 (4.4) | -9.5 (10.6) | -4.3 (5.7) | 0.5 (7.7) | -9.0 (12.7) | -1.5 (4.7)
  Change from BL at 24h post dose | -2.2 (3.3) | -3.7 (8.5) | -4.5 (8.4) | -4.3 (2.6) | -7.0 (3.5) | -6.5 (3.0) | -4.3 (4.9) | -5.5 (8.9) | 0.0 (0.0) | -2.0 (2.8)
  Change from BL at FU | -5.5 (4.9) | -1.3 (7.4) | -5.0 (4.3) | -7.3 (2.2) | -11.0 (5.3) | -3.0 (9.3) | -9.8 (4.9) | -7.0 (2.6) | -16.0 (14.1) | -3.5 (5.0)

92. Primary Outcome: SAD: Change From Baseline in ECG Results by Time Point: QRS Interval
Description: as for outcome 91
Time Frame: Pre-dose, Day 1, Day 7
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SAD Group I Placebo | SAD Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group II 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
msec
  Baseline (Pre-dose Day 1) | 103.0 (8.3) | 97.0 (9.6) | 99.3 (3.3) | 97.8 (7.6) | 106.5 (10.2) | 92.5 (13.9) | 104.5 (10.6) | 94.0 (8.8) | 95.0 (7.1) | 105.5 (8.3)
  Change from baseline at 1h | -0.7 (2.0) | 1.0 (5.2) | -1.3 (0.5) | 0.3 (2.2) | 0.0 (2.8) | 3.5 (3.4) | 1.5 (6.4) | 26.0 (6.9) | 1.0 (1.4) | 0.0 (2.8)
  Change from BL at 2h post dose | -2.0 (3.0) | 0.7 (3.2) | -1.3 (1.3) | -0.3 (1.0) | -2.5 (1.0) | 3.0 (2.6) | 2.5 (7.2) | 20.5 (7.7) | 0.0 (0.0) | -2.0 (2.8)
  Change from BL at 4h post dose | -1.0 (3.0) | -0.7 (2.2) | -1.3 (1.7) | -0.8 (0.5) | -2.0 (0.0) | 2.0 (2.8) | 2.5 (3.0) | 17.0 (6.0) | 0.0 (2.8) | -3.5 (3.4)
  Change from BL at 6h post dose | 0.3 (3.8) | 0.3 (1.6) | 0.8 (2.6) | -0.3 (2.8) | -1.5 (1.0) | 3.5 (2.5) | 1.5 (2.5) | 14.5 (5.3) | 1.0 (1.4) | -1.5 (3.4)
  Change from BL at 8h post dose | -2.0 (2.8) | -1.0 (1.3) | 1.3 (3.3) | -0.8 (2.1) | -2.0 (1.6) | 2.5 (1.9) | 0.0 (6.7) | 13.0 (4.8) | 0.0 (0.0) | -0.5 (1.9)
  Change from BL at 12h post dose | -0.7 (3.6) | -1.7 (1.0) | 0.3 (2.5) | -0.3 (2.5) | -1.5 (2.5) | 1.0 (2.6) | 2.5 (3.0) | 7.0 (2.0) | 0.0 (0.0) | -2.5 (3.0)
  Change from BL at 24h post dose | -2.7 (5.3) | -1.7 (3.4) | -1.3 (0.5) | -2.3 (2.2) | -1.5 (1.9) | 1.5 (4.4) | 0.0 (1.6) | 4.0 (0.0) | -3.0 (4.2) | -1.0 (2.0)
  Change from BL at FU | -1.3 (6.2) | -0.7 (4.4) | -1.3 (3.5) | 0.8 (6.4) | -2.5 (4.1) | 0.0 (3.3) | -3.0 (5.3) | -0.5 (2.5) | -1.0 (4.2) | -1.5 (4.7)

93. Primary Outcome: SAD: Change From Baseline in ECG Results by Time Point: QT Interval
Description: as for outcome 91
Time Frame: Pre-dose, Day 1, Day 7
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SAD Group I Placebo | SAD Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group II 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 2 | 4
msec
  Baseline (Pre-dose Day 1) | 400.0 (18.6) | 415.0 (23.5) | 393.3 (15.4) | 416.0 (15.6) | 404.0 (11.4) | 409.0 (28.2) | 396.3 (15.9) | 398.3 (17.3) | 373.0 (7.1) | 396.0 (12.8)
  Change from baseline at 1h | 9.7 (12.7) | -4.3 (13.6) | 2.3 (6.4) | -8.5 (9.5) | 10.5 (5.3) | -3.0 (7.4) | -5.8 (17.6) | 8.8 (22.7) | -11.0 (1.4) | -15.5 (14.3)
  Change from BL at 2h post dose | 3.0 (8.5) | -7.3 (16.2) | 4.8 (21.4) | 0.5 (9.7) | 9.0 (10.9) | -2.5 (6.6) | 3.3 (17.1) | 4.8 (21.9) | -2.0 (5.7) | 16.0 (11.7)
  Change from BL at 4h post dose | 9.3 (7.5) | -3.7 (16.9) | 3.3 (9.0) | 6.0 (7.1) | 7.0 (12.9) | -2.0 (11.4) | -3.8 (16.7) | 1.8 (14.6) | 7.0 (4.2) | -4.0 (8.5)
  Change from BL at 6h post dose | -6.7 (8.8) | -16.0 (14.8) | -9.8 (8.5) | -19.5 (7.4) | -3.5 (13.2) | -11.0 (6.2) | -19.3 (9.2) | -4.8 (16.3) | -14.0 (5.7) | -13.0 (8.4)
  Change from BL at 8h post dose | -8.7 (4.4) | -24.0 (9.9) | -6.8 (9.1) | -18.5 (4.0) | -4.0 (16.6) | -16.0 (9.8) | -14.8 (9.3) | -5.3 (7.1) | -17.0 (15.6) | -9.0 (9.3)
  Change from BL at 12h post dose | -8.7 (3.3) | -24.3 (16.3) | -2.8 (9.0) | -15.5 (11.2) | -6.5 (13.0) | -22.5 (6.8) | -12.3 (7.5) | -13.3 (15.9) | -18.0 (17.0) | -10.0 (15.5)
  Change from BL at 24h post dose | -6.7 (6.1) | -23.0 (13.5) | -11.8 (3.0) | -15.5 (16.5) | -4.5 (8.2) | -17.0 (14.7) | -10.3 (13.3) | 2.3 (4.9) | -3.0 (18.4) | -7.0 (3.8)
  Change from BL at FU | -12.0 (4.3) | -18.3 (11.4) | -13.8 (6.7) | -12.5 (9.8) | -9.0 (5.0) | -12.0 (13.4) | -8.3 (12.4) | -7.8 (10.1) | -2.0 (25.5) | -1.0 (8.9)

94. Primary Outcome: SAD: Change From Baseline in ECG Results by Time Point: QTcB Interval
Description: as for outcome 91
Time Frame: Pre-dose, Day1, Day 7
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: msec
Groups:
- SAD Group I Placebo: SAD group I Placebo
- SAD Group II Placebo: SAD group II Placebo
Arm/Group | SAD Group I Placebo | SAD Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group II 100mg + Food
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 2
msec
  Baseline (Pre-dose Day 1) | 379.3 (21.0) | 385.5 (9.8) | 382.0 (21.4) | 390.5 (8.9) | 383.8 (24.8) | 386.3 (8.0) | 382.0 (10.9) | 378.5 (19.1) | 367.5 (24.7) | 382.3 (22.0)
  Change from BL at 1h | 1.7 (7.7) | -0.7 (10.1) | -1.0 (2.8) | -0.3 (6.7) | -3.5 (5.0) | 1.8 (7.3) | 3.0 (8.6) | 39.0 (19.0) | 12.5 (29.0) | 16.0 (7.9)
  Change from BL at 2h post dose | -0.5 (12.8) | -2.8 (9.3) | -4.0 (18.2) | -6.5 (7.9) | -10.8 (9.6) | 3.0 (8.4) | 9.8 (8.3) | 41.3 (21.7) | 4.5 (25.3) | 10.3 (4.0)
  Change from BL at 4h post dose | 5.5 (15.2) | -1.5 (17.1) | -7.3 (3.3) | -8.3 (11.9) | -1.5 (7.0) | 6.0 (17.8) | 6.5 (6.2) | 38.5 (10.7) | 9.0 (28.3) | 1.8 (8.2)
  Change from BL at 6h post dose | 12.7 (4.8) | 3.7 (8.4) | 11.5 (5.8) | 4.0 (13.1) | 0.0 (14.9) | 14.0 (11.0) | 17.8 (1.0) | 41.8 (13.8) | 20.0 (15.6) | 15.5 (6.6)
  Change from BL at 8h post dose | 3.0 (12.3) | 1.2 (9.3) | -4.8 (7.8) | 6.8 (14.2) | 8.5 (18.7) | 5.5 (12.1) | 8.0 (7.4) | 37.5 (19.3) | 5.0 (12.7) | 5.0 (6.5)
  Change from BL at 12h post dose | 7.0 (8.3) | 3.8 (8.9) | -1.0 (2.2) | -2.8 (14.0) | 2.8 (13.0) | 11.5 (13.1) | 17.8 (5.2) | 36.0 (9.4) | 17.5 (2.1) | 9.5 (10.3)
  Change from BL at 24h post dose | 11.7 (19.3) | 0.0 (8.6) | 0.0 (11.3) | 0.8 (15.1) | 3.0 (7.1) | 1.5 (6.5) | 5.3 (9.0) | 15.8 (4.9) | -0.5 (21.9) | -2.5 (5.7)
  Change from BL at FU | 5.3 (17.6) | 13.0 (15.4) | 4.8 (18.8) | 10.8 (15.9) | 8.3 (19.8) | 13.3 (12.7) | -3.5 (6.5) | 9.0 (14.4) | 9.0 (28.3) | 9.8 (18.5)

95. Primary Outcome: Terminal Elimination Half-life (T1/2) of KH176 Over 24 Hours: SAD
Description: Plasma concentrations of KH176 were analysed after single dose administration of doses 10mg, 30mg, 100mg (with and without food), 300mg, 800mg, 2000mg b.i.d.
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
hours | 0 (0) | 10.3 (14.6) | 9.10 (15.2) | 9.64 (4.29) | 9.80 (19.1) | 11.5 (4.73) | 9.09 (3.83)

96. Primary Outcome: Terminal Elimination Half-life (T1/2) of KH183: SAD
Description: Plasma concentrations of KH183 were analysed after single dose administration of doses 10mg, 30mg, 100mg (with and without food) , 300mg, 800mg, 2000mg b.i.d.
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
hours | 16.6 (5.86) | 17.8 (19.0) | 15.4 (8.44) | 14.3 (18.9) | 17.2 (18.5) | 18.9 (18.7) | 14.9 (7.86)

97. Primary Outcome: Maximum Concentration (Cmax) of KH176: SAD Group
Description: as for outcome 95
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
ng/mL | 12.9 (21.3) | 56.2 (21.0) | 167 (27.2) | 766 (53.9) | 2170 (27.9) | 5990 (20.9) | 165 (7.40)

98. Primary Outcome: Maximum Concentration (Cmax) of KH183 Over 24 Hours: SAD
Description: as for outcome 96
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
ng/mL | 14.2 (49.5) | 49.4 (9.00) | 168 (29.6) | 497 (17.6) | 1100 (9.58) | 1780 (26.3) | 117 (20.0)

99. Primary Outcome: Maximum Concentration (Cmax) of KH183 (Active Metabolite of KH176): MAD Group
Description: Plasma concentrations of KH183 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.: Cmax was obtained directly from the concentration-time data.
Time Frame: Predose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cmax Dose 100mg: Maximum concentration - 100mg
- Cmax - Dose 200mg: Maximum concentration - 200 mg
- Cmax - Dose 400mg: Maximum concentration - 400mg
Arm/Group | Cmax Dose 100mg | Cmax - Dose 200mg | Cmax - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  Day 1 | 99.4 (20.9) | 251 (18.0) | 550 (14.1)
  Day 7 | 152 (37.5) | 250 (10.6) | 450 (28.3)

100. Primary Outcome: Maximum Concentration (Cmax) of KH176: MAD
Description: Plasma concentrations of KH176 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: pre-dose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cmax Dose 100mg | Cmax - Dose 200mg | Cmax - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  Day 1 | 184 (57.0) | 313 (20.0) | 1330 (27.3)
  Day 7 | 353 (19.1) | 748 (29.3) | 2100 (27.2)

101. Primary Outcome: Time to Maximum Concentration (Tmax) of KH176 Over 24 Hours: SAD
Description: as for outcome 95
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
hours | 1.03 (55.5) | 1.03 (55.5) | 0.931 (83.4) | 1.10 (85.6) | 1.36 (20.5) | 0.931 (102) | 2.45 (23.7)

102. Primary Outcome: Time to Reach Peak Plasma Concentration (Tmax) of KH183: SAD
Description: Plasma concentrations of KH183 were analysed after single dose administration of doses 10mg, 30mg, 100mg (with and without food), 300mg, 800mg, 2000mg b.i.d.
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
ng/mL | 1.32 (34.8) | 1.46 (29.1) | 1.32 (34.8) | 1.31 (34.7) | 1.61 (14.5) | 1.57 (33.7) | 2.45 (23.7)

103. Primary Outcome: Time to Maximum Concentration (Tmax) of KH176 at Day 1, Day 7: MAD Group
Description: Plasma concentrations of KH176 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: pre-dose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Tmax Dose 100mg: Time to Maximum concentration - 100mg
- Tmax - Dose 200mg: Time to Maximum concentration - 200 mg
- Tmax - Dose 400mg: Time to Maximum concentration - 400mg
Arm/Group | Tmax Dose 100mg | Tmax - Dose 200mg | Tmax - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
hours
  Day 1 | 1.57 (173) | 1.73 (16.7) | 0.866 (70.4)
  Day 7 | 0.931 (48.1) | 1.86 (14.5) | 1.36 (85.5)

104. Primary Outcome: Time to Maximum Concentration (Tmax) of KH183 (Active Metabolite of KH176): MAD Group
Description: Plasma concentrations of KH183 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.. tmax was obtained directly from the concentration-time data.
Time Frame: Predose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tmax Dose 100mg | Tmax - Dose 200mg | Tmax - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
hours
  Day 1 | 2.06 (116) | 1.57 (33.7) | 1.22 (23.7)
  Day 7 | 1.19 (36.6) | 1.46 (29.1) | 1.61 (48.1)

105. Primary Outcome: Accumulation Factor (Racc) of KH176 Over 7 Days: MAD Group
Description: Plasma concentrations of KH176 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.. Racc was calculated as follows: AUCtau day 7/ AUCtau day 1.
Time Frame: Pre-dose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Racc Dose 100mg: Accumulation factor - 100mg
- Racc- Dose 200mg: Accumulation factor - 200 mg
- Racc - Dose 400mg: Accumulation factor - 400mg
Arm/Group | Racc Dose 100mg | Racc- Dose 200mg | Racc - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
ratio | 2.52 (31.2) | 2.65 (2.5) | 2.17 (14.4)

106. Primary Outcome: Accumulation Factor (Racc) of KH183 (Active Metabolite of KH176): MAD Group
Description: Plasma concentrations of KH183 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.: Accumulation factor was calculated as follows: AUCtau day 7/ AUCtau day 1.
Time Frame: Predose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set. The placebo subjects were excluded from the PK analysis per-protocol set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Racc Dose 100mg | Racc- Dose 200mg | Racc - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
ratio | 1.86 (46.7) | 1.32 (13.1) | 1.19 (24.7)

107. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUClast) of KH183: SAD Group
Description: as for outcome 96
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
h*ng/mL | 151 (26.7) | 547 (12.4) | 1810 (37.4) | 4830 (11.8) | 11700 (20.2) | 23900 (22.2) | 1590 (26.1)

108. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUClast) of KH176: SAD Group
Description: as for outcome 95
Time Frame: pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
h*ng/mL | 75 (14.8) | 389 (8.16) | 1310 (16.7) | 6320 (20.2) | 21000 (27.5) | 61200 (9.07) | 1650 (1.67)

109. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUCtau) of KH176: MAD Group:
Description: Plasma concentrations of KH176 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: Pre-dose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- AUCtau Dose 100mg: Area under the plasma concentration-time curve during a dose interval- 100mg
- AUCtau - Dose 200mg: Area under the plasma concentration-time curve during a dose interval - 200 mg
- AUCtau - Dose 400mg: Area under the plasma concentration-time curve during a dose interval - 400mg
Arm/Group | AUCtau Dose 100mg | AUCtau - Dose 200mg | AUCtau - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
h*ng/mL
  Day 1 | 1090 (49.3) | 2250 (26.1) | 6890 (19.2)
  Day 7 | 2760 (22.6) | 5960 (26.8) | 14900 (28.2)

110. Primary Outcome: Area Under the Plasma Concentration-time Curve During a Dose Interval (AUCtau) of KH183 (Active Metabolite of KH176): MAD Group
Description: Plasma concentrations of KH183 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: Predose at Day 1, 2, 4, 7, and post-dose at Day 1 and Day 7 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
Population: Per protocol set. The placebo subjects were excluded from the PharmaocoKinetics (PK) analysis per-protocol set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | AUCtau Dose 100mg | AUCtau - Dose 200mg | AUCtau - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
h*ng/mL
  Day 1 | 702 (29.2) | 1680 (21.0) | 3600 (11.1)
  Day 7 | 1310 (29.5) | 2220 (12.7) | 4270 (30.5)

111. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Until Infinity (AUCl0-inf) of KH183: SAD
Description: as for outcome 96
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
h*ng/mL | 234 (26.7) | 881 (19.6) | 2690 (38.4) | 6690 (11.0) | 18700 (26.7) | 41300 (10.5) | 2410 (29.1)

112. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Until Infinity (AUCl0-inf) of KH176: SAD
Description: Plasma concentrations of KH176 were analysed after single dose administration of doses 10mg, 30mg, 100mg (with and without food) , 300mg, 800mg, 2000mg b.i.d.
Time Frame: Pre-dose (5 min before dosing) and 0.5, 1, 1.5, 2, 3, 6, 8, 12, and 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I 100mg + Food
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4
h*ng/mL | 0 (0) | 474 (8.39) | 1540 (13.1) | 7500 (19.1) | 25800 (33.9) | 79100 (8.82) | 1970 (1.04)

113. Primary Outcome: KH176: Percentage of Administered Dose Excreted in Urine: SAD
Description: Urine concentrations of KH176 were analysed after single dose administration of doses 10mg, 30mg, 100mg (with and without food), 300mg, 800mg, 2000mg b.i.d.
Time Frame: 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 4 | 4
percentage of dose excreted | 9.71 (37.4) | 10.5 (45.6) | 10.4 (29.5) | 9.53 (65.2) | 10.9 (41.6) | 12.4 (20.7)

114. Primary Outcome: KH183: Percentage of Administered Dose Excreted in Urine: SAD
Description: as for outcome 113
Time Frame: 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 4 | 4
percentage of dose excreted | 4.56 (53.0) | 6.42 (14.5) | 5.18 (28.8) | 3.81 (82.9) | 3.86 (31.0) | 3.33 (32.8)

115. Primary Outcome: KH176 + KH183: Percentage of Administered Dose Excreted in Urine: SAD
Description: as for outcome 113
Time Frame: 24 hours post-dose
Population: Per protocol set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted
Arm/Group | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 4 | 4
percentage of dose excreted | 14.4 (40.0) | 17.2 (28.6) | 15.8 (24.5) | 13.4 (69.9) | 14.8 (38.4) | 15.9 (16.4)

116. Primary Outcome: KH176: Percentage of Administered Dose Excreted in Urine: MAD
Description: Urine concentrations of KH176 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: Day 7 post dose
Population: Per protocol set. The placebo subjects were excluded from the Pharmacokinetics (PK) analysis per-protocol set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted
Groups:
- MAD Group Dose 100mg: 100mg KH176 - Multiple dose: Percentage of administered dose excreted
- MAD Group - Dose 200mg: 200mg KH176 - Multiple dose: Percentage of administered dose excreted
- MAD Group - Dose 400mg: 400mg KH176 - Percentage of administered dose excreted
Arm/Group | MAD Group Dose 100mg | MAD Group - Dose 200mg | MAD Group - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
percentage of dose excreted | 14.9 (77.8) | 13.4 (36.4) | 14.0 (14.5)

117. Primary Outcome: KH183: Percentage of Administered Dose Excreted in Urine: MAD
Description: Urine concentrations of KH183 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: Post dose Day 7
Population: Per protocol set. The placebo subjects were excluded from the Pharmacokinetics (PK) analysis per-protocol set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted
Arm/Group | MAD Group Dose 100mg | MAD Group - Dose 200mg | MAD Group - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
percentage of dose excreted | 5.30 (120.2) | 3.79 (39.2) | 4.85 (43.8)

118. Primary Outcome: KH173 + KH183: Percentage of Administered Dose Excreted in Urine: MAD
Description: Urine concentrations of KH176 and KH183 were analysed after multiple-dose administration of doses of 100, 200 and 400 mg b.i.d.
Time Frame: Day 7 Post dose
Population: Per protocol set. The placebo subjects were excluded from the Pharmacokinetics (PK) analysis per-protocol set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose excreted
Arm/Group | MAD Group Dose 100mg | MAD Group - Dose 200mg | MAD Group - Dose 400mg
Number analyzed (Participants) | 4 | 4 | 4
percentage of dose excreted | 20.7 (79.3) | 17.4 (33.3) | 19.0 (17.9)

ADVERSE EVENTS:
Groups:
- Placebo: Placebo
Arm/Group | Group I Placebo | Group II Placebo | SAD Group I 10mg | SAD Group II 30mg | SAD Group I 100mg | SAD Group II 300mg | SAD Group I 800mg | SAD Group II 2000mg | Group I Placebo + Food | Group I 100mg + Food | MAD Group III 200mg | MAD Group IV 400mg | MAD Group V 800mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 2/4 | 3/4 | 4/4 | 1/4 | 0/4 | 4/4 | 1/2 | 1/4 | 3/4 | 3/4 | 4/4 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I Placebo (N=6) | Group II Placebo (N=6) | SAD Group I 10mg (N=4) | SAD Group II 30mg (N=4) | SAD Group I 100mg (N=4) | SAD Group II 300mg (N=4) | SAD Group I 800mg (N=4) | SAD Group II 2000mg (N=4) | Group I Placebo + Food (N=2) | Group I 100mg + Food (N=4) | MAD Group III 200mg (N=4) | MAD Group IV 400mg (N=4) | MAD Group V 800mg (N=4) | Placebo (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depersonalisation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Dysgeusia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 3 (5)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No